## Official Study Title: Effects of Dehydroepiandrosterone in Pulmonary Hypertension

Document: Protocol

NCT Number: NCT03648385

Document Date: August 12, 2021

## Research Strategy A. Significance

**A1. Sexual dimorphism in PH prevalence and outcomes.** Female sex is the strongest clinical risk factor for PAH, with a 4:1 female-to-male ratio reported from the largest registry.<sup>31</sup> Despite the increased risk of PAH in women, women with PAH have better survival than men.<sup>1,32</sup> RV function is an important cause of morbidity and mortality in PAH as well as highly prevalent heart and lung disease but determinants of the RV response are entirely unknown.<sup>7-9</sup> We and others have shown that female sex is associated with better RV systolic function in both health and disease, including PAH and left heart failure.<sup>2,33-35</sup> Targeted PAH therapy leads to greater improvements in RVEF (demonstrated after just several months of treatment) in women as compared to men and partially explains better outcomes in women.<sup>4,36</sup> Demonstration that DHEA has direct RV and sexbased effects will support the hypothesis that sex hormones play an important role in disease pathogenesis and provide insight into sex hormone manipulation as a treatment strategy in PAH.

**A2. Beneficial effects of DHEA on pulmonary vasculature.** DHEA and DHEA-S are precursors in the biosynthesis of androgens and estrogens (Figure 2), but <u>we and others have shown biological effects of DHEA which are independent of other sex hormones.</u> As PAH is more common in women than in men, estrogen has been implicated as a mechanistic factor in disease development and in fact estrogen can induce PH in some animal models. In contrast, DHEA appears to be consistently beneficial in experimental PH via mechanisms which are entirely independent of E2 signaling (Table 1), although these studies have been

done predominantly in male animals (as with most published studies in animal models for PH). 16-20, 39 In humans, lower DHEA-S levels have been linked to systemic endothelial dysfunction and track independently with flow mediated dilatation; these effects can be rescued with DHEA supplementation. 41, 42 A recent study of unbiased metabolomic profiling demonstrated DHEA-S and its metabolites were reduced in PAH patients compared to healthy controls; lower circulating levels of DHEA-S were associated with mortality in PAH. 14

Pregnenolone

Progesterone

Androstenedione

Estradiol

Estrone

Figure 2. Sex hormone synthesis

Table 1. Experimental data supporting beneficial effects of DHEA

| Model | DHEA Effects | Proposed Mechanism |
|---|---|---|
| | Prevent, rescue PH | BK <sub>Ca</sub> channels <sup>16, 17</sup> |
| Hypoxia | Rescue PH | BK <sub>Ca</sub> , inhibits 5HT-, KCl-induced SMC growth <sup>37</sup> |
| | Rescue RV | Reduces cardiomyocyte proliferation <sup>18</sup> |
| Altitude | Prevent, rescue PH | sGC <sup>38</sup> |
| MCT, Prevent, rescue PH | | Inhibits Src, STAT3, Pim1 |
| PASMCs | | Increases BMPR2, miR-204 <sup>20</sup> |
| MCT-PNX | Prevent, rescue | Inhibits RhoA/Rho kinase 39 |
| SU5416/ | Rescue RV>PH | Reduces RV capillary rarefaction, |
| Hypoxia | Rescue RV>PH | apoptosis, ROS via STAT3 19 |
| | Antichronotropic, | Reduces T-type Ca channels <sup>22</sup> |
| Cardiomyocytes | Antihypertrophic | Inhibits natriuretic peptide |
| | Antihypertrophic | Reduces ET-1 induced hypertrophy <sup>21</sup> Inhibits BNP |

BK<sub>Ca</sub>=large conductance Ca<sup>2+</sup> activated K channel; 5HT=serotonin; SMC=smooth muscle cell; STAT3=signal transducer and activator of transcription 3; BMPR2=bone morphogenetic receptor type II; MCT=monocrotaline; PNX=pneumonectomy

# **A3. DHEA and cardiac function.** Low DHEA-S levels have been associated

with an increased risk of death in heart disease, cardiac allograft vasculopathy, and heart failure severity. 43-47 DHEA reverses cardiomyocyte hypertrophy induced by ET-121 and prevents myocardial fibrosis and contractile dysfunction by restoring oxidative balance, mitigating the actions of AGE products and its receptors, and improving tissue levels of collagen and fibronectin. 48, 49 Myocardial fibrosis is a key phenotypic change in RV remodeling and decompensation in PAH. 50 DHEA treatment improves cardiac index and inhibits RV capillary rarefaction, fibrosis, and oxidative stress, suggesting an RV-disproportionate or -specific effect. While first established as major regulators of pulmonary vascular tone, NO and ET-1 also influence RV phenotype. There is a DHEA receptor coupled to endothelial NO synthase (eNOS) and DHEA regulates ET-1 synthesis and inhibits ET-1 promoter activity. Our data show a definitive link between lower DHEA-S levels, PAH and RV function in men and women (Section C3), independent of E2. DHEA's key links with RV remodeling, NO and ET-1 could explain sex-based differences in outcomes and PAH therapeutic response (Figure 1). If we see that DHEA effects RV function, we will next validate these findings in a multicenter, parallel arm, Phase II RCT.

**A4.** Important markers of RV phenotype and oxidative stress. The RV as compared to the left ventricle (LV) has complex rotational motion from a unique myocardial fiber arrangement requiring highly sensitive methods to detect conformational changes. RV metrics obtained by cardiac MRI are highly accurate and MRI is the gold standard for RV assessment. 52-55 **Longitudinal strain**, which is an angle-independent method of assessing RV systolic function measured by echocardiography is associated with survival in PAH and tracks with PAH therapy. 56, 57 Echocardiography is inferior to MRI, however, and pixel based multimodality tissue

tracking (MTT) using MRI cine images is now available to quantify strain. This method has been described in PAH (Figure 3) and is highly reproducible, with intra- and inter-observer mean differences of -0.5 ± 1.5% and -0.6 ± 2.1% respectively. Security Assessment of strain by MRI appears highly sensitive for the detection of early pre-clinical changes in RV contractility, making this an ideal primary end point to detect an efficacy signal in this "proof of concept" study. RVEF is a key determinant of outcome in RV failure regardless of etiology including PAH. Per RVEF predicts outcome in PAH and changes in RV measures track with even short-term (<1 hour, typically several months) exposure to PAH therapies. A 36, 59-61



**Galectin-3**, a marker of myocardial extracellular matrix metabolism and fibrosis, is elevated in the plasma of PAH patients<sup>62</sup> and inversely correlates with MRI-based measures including RVEF.<sup>63</sup> **RAGE** levels are elevated in plasma and explanted lungs of PAH patients.<sup>64, 65</sup> RAGE is a strong STAT3 activator (key in PAH pathophysiology and one of the mechanisms by which DHEA reverses experimental PH).<sup>20, 65</sup> Soluble RAGE has been shown to inhibit myocardial apoptosis via STAT3 activation in cardiac ischemia/reperfusion injury.<sup>66</sup> While **oxidative stress** is challenging to quantify in patients, we propose measuring the levels of MPO, a major source of ROS linked to systemic inflammation with a track record in cardiovascular disease as a redox biomarker,<sup>67-69</sup> and sNOX2-dp, a marker of NADPH oxidase activity, which predicts microvascular obstruction in coronary disease.<sup>70-72</sup>

**A5. DHEA's efficacy in clinical trials and evidence of safety.** Most RCTs of DHEA have been conducted in adrenal insufficiency and systemic lupus erythematosus. No serious side effects were reported in these RCTs including >1200 patients, with reversible mild androgenic side effects (oily skin, hirsutism, acne) in some studies.<sup>73-75</sup> DHEA 50 mg daily improved systemic vascular stiffness and reduced interleukin (IL)-6 as well as tumor necrosis factor-α in healthy adults <sup>76</sup>, cytokines implicated in PAH pathogenesis and associated with symptoms and survival in PAH<sup>77, 78</sup>. In eight patients with PH related to COPD, treatment with three months of DHEA was associated with a significant increase in six-minute walk distance (6MWD) and improvements in hemodynamics without adverse effects.<sup>79</sup> While this small study is promising, it was uncontrolled, open-label, and did not include patients with PAH. We have studied anastrozole as an approach to reducing E2 levels in PAH (Section C4). There was no effect on DHEA-S levels<sup>15</sup>, so that the observed reductions in E2 and increase in 6MWD were unrelated to DHEA. Furthermore, our preliminary data show that DHEA is linked to the risk of more severe disease independent of changes in E2 and other hormones. Considering the consistently favorable findings in experimental and human PAH and the low risk of the intervention, there is a strong scientific premise and critical need for a clinical trial examining DHEA in the treatment of PAH.

**A6. DHEA** alters phenotype of cultured endothelial cells. DHEA at variable concentrations (10<sup>-5</sup>–10<sup>-8</sup> M) induces changes in human endothelial cell phenotype. <sup>20, 80-84</sup> Effects include enhanced eNOS expression and NO synthesis and modulated ET-1 secretion. <sup>24, 82</sup> DHEA reduces inflammatory signaling implicated in atherosclerosis in human systemic vein endothelial cells. <sup>80, 84</sup> Human PAECs actively metabolize DHEA and treatment of PAECs from PAH patients decreases STAT3 activation, <sup>20, 85</sup> an important mediator of pulmonary vascular remodeling. The effect of DHEA treatment on pulmonary endothelial NO and ET-1 synthesis in PAH has not been studied nor has the effect of patient sex on PAEC response to DHEA treatment.

A7. Intersection of sex and sex hormones with key mechanistic pathways in PAH and the RV. Extensive data from preclinical models have implicated sex hormones in PH but translation of these findings to human PAH has lagged behind. We (and others) have recently shown that men with PAH have worse hemodynamics as compared to women with PAH<sup>5, 86</sup> and that sex hormone levels as well as genetic variants in hormone pathways are linked to PAH risk and RV morphology.<sup>2, 87, 88</sup> Men with PAH are more likely to respond to PDE5i (a major class of PAH treatment), while women with PAH respond better to ERAs (another widely used therapy) than men.<sup>3, 6</sup> Differential responses to therapy may be due to the interaction of key mechanistic pathways in PAH with DHEA (Figure 1). Women have greater levels of NO biosynthesis compared to men, while men have higher levels of ET-1 and greater ET-1-mediated vasconstriction.<sup>25, 27, 29</sup> Sex hormones directly modulate NO/cyclic guanosine monophosphate (cGMP) signaling and circulating ET-1 levels.<sup>28, 89, 90</sup> Animal models of PH have increased female penetrance and show detrimental effects of E2 on the pulmonary vasculature under some but not all conditions.<sup>91-94</sup> Unlike E2, which has conflicting and paradoxical effects on cardiopulmonary function, DHEA shows consistently beneficial effects on the pulmonary vasculature and the

**A8. Critical need to improve treatment of PAH.** PAH treatment is extremely expensive <sup>95, 96</sup> and annual medication costs exceed \$200,000. While a recent trial suggests a benefit of up-front combination treatment with PDE5i and ERA<sup>3, 6, 97</sup>, it is possible that the combination approach simply assures a greater proportion of individuals receive the most effective drug for their sex or hormonal milieu. Understanding treatment response heterogeneity is critical for cost containment and for the advancement of precision medicine in PAH. If we show sex-based differential responses to DHEA (*in vivo* or in PAECs *in vitro*), this will inform our understanding of why treatment responses with PAH therapies differ by sex and allow for the adaptive design of future RCTs.

**A9. Scientific Premise.** Preclinical and limited human studies indicate that DHEA favorably impacts endothelial cell-derived vasoactive mediators and myocardial remodeling. We have shown that men and women with PAH have lower levels of DHEA-S and that low levels predict more severe disease independent of E2 levels (Section C3); a recent study linked low DHEA-S levels to mortality in PAH. Therefore, there is a need for determining the safety and efficacy of DHEA in humans with PAH. Only an interventional study with a complementary cell based aim can untangle the role of DHEA in cardiopulmonary function in PAH.

#### **B.** Innovation

#### **Conceptual Innovation:**

- We will test the idea that DHEA, an endogenous hormone, alters RV and endothelial phenotype in PAH.
- Restoration of low DHEA levels may correct the derangements that lead to PAH and have direct effects on RV adaptation rather than simply combating vasoconstriction as is the case for all currently available pulmonary vasodilators.
- DHEA is an inexpensive and safe supplement not previously studied in human PAH and RV failure that has effects independent of those of other sex hormones, like E2.
- These studies will have implications for precision care in PAH in that already available therapies may be preferentially advised based on an individual's sex or sex hormone milieu. Our objectives for this proposal and beyond are well-aligned with the NIH Strategic Plan for Lung Vascular Research<sup>98</sup> and a recent workshop on enhancing treatments for PAH through precision medicine.<sup>99</sup>

#### **Technical Innovation:**

- To our knowledge, there are no RCTs of this size in PAH with the primary end point of MRI-derived RVEF the proximate cause of death in PAH and PH for which there are no approved therapies.
- The use of a cross-over design with carefully chosen end points to capture RV phenotype (imaging, markers
  of RV fibrosis and oxidative stress), known major mechanistic mediators in PAH (NO and ET-1), as well as
  common intermediate end points in PAH (6MWT, health-related quality of life [HRQOL], functional class) will
  maximize precision, minimize within subject variability, and allow for robust patient-level analyses to detect
  variable signals based on an

individual's sex, age, race/ethnicity, and PAH sub-type.

 Mechanistic studies of DHEA's effects will use PAECs isolated from PAH patients, a very novel approach.

 Table 2. Sex related differences in hemodynamic values in 1211 PAH patients

| Variable | Age | Difference, men<br>and women | 95% CI | P value |
|---|---|---|---|---|
| RAP, mm Hg | • | 1.36 | 0.44 - 2.27 | 0.004 |
| mPAP, mm Hg | < 45 | 5.43 | 2.20 - 8.66 | 0.001 |
| | 45-54 | 1.37 | <b>-</b> 2.64 – 5.37 | 0.50 |
| | 55-64 | -1.45 | <b>-</b> 5.70 <b>–</b> 2.81 | 0.50 |
| | 65+ | 3.06 | -1.31 – 7.43 | 0.17 |
| Cardiac output, L/min | | -0.21 | -0.43 - 0.01 | 0.06 |
| PVR, Wood units | | 1.23 | 0.18 - 2.27 | 0.02 |

Adjusted for age (if no sex\*age interaction), race, height, weight, study

#### C. Approach

C1. Men have worse disease than women with PAH. First, we determined whether men and women have baseline

differences that may explain distinct PAH epidemiology and outcomes. In a large (n = 1211), pooled analysis of patient-level data from Phase III RCTs in PAH submitted to the FDA, men with PAH had higher right atrial pressure (RAP) and pulmonary vascular resistance (PVR) compared to women with PAH (Table 2). Younger men had higher mean pulmonary artery pressures (mPAP) than younger women.

**C2. Sex hormones and RV function.** We next sought to determine whether sex hormone levels are associated with RV function as an explanation for dimorphic outcomes in PAH. We examined sex hormone levels from a large (n = 3695) cardiovascular disease-free cohort (Multi-Ethnic Study of Atherosclerosis [MESA]) generalizable to RV failure irrespective of cause.<sup>2, 100</sup> Higher levels of DHEA were associated with lower RVEF (calculated from RV stroke volume/RV end-diastolic volume), higher RV stroke volume (calculated from RV end-diastolic – RV end-systolic volume), and larger RV end-diastolic volume in healthy post-

menopausal women. While a lower RVEF and larger RV stroke volume seem difficult to reconcile, higher (but not necessarily detrimental) RV end-diastolic volume with increasing DHEA levels would result in larger RV

stroke volume (which may be beneficial) and numerically but not necessarily pathologically lower RVEF. In fact, virtually all participants had a normal RVEF in MESA as these are "disease-free" adults. Our data in patients with PAH show that higher DHEA-S levels protect against PAH and improve RV function (Section C3), apparently contradicting the MESA findings. These inconsistencies likely result from the measurement of DHEA-S (in PAH) versus DHEA (in MESA)(the former having more stability), studying a diseased versus a healthy population, and the analysis of DHEA's cross-sectional associations with normal RV indices in MESA. The only way to answer these questions is an interventional study of DHEA in PAH as proposed.



C3. DHEA in human PAH.

Given our observations in healthy participants from MESA, we studied whether DHEA and other sex hormones were risk factors for PAH in men<sup>101</sup> and women. We included 23 men with PAH matched by age and body mass index

Table 3. Lower DHEA-S levels and markers of disease severity in men and women with PAH

| | | Men | | Women | | |
|---|---|---|---|---|---|---|
| Variable | Estimate | 95% CI | P value | Estimate | 95% CI | P value |
| 6MWD, m | -6.1 | -47.1, 34.9 | 0.750 | -30.2 | -54.0, -6.5 | 0.013 |
| RAP, mm Hg | 2.7 | -0.6, 4.8 | 0.020 | 1.6 | 0.3, 2.8 | 0.019 |
| mPAP, mm Hg | 0.0 | -5.4, 5.3 | 0.999 | 3.6 | 1.8, 5.4 | <0.001 |
| Cardiac output, L/min | -0.6 | -1.4, 0.2 | 0.140 | -0.2 | -0.4, 0.0 | 0.067 |
| PVR, Wood units | 3.4 | 0.9, 5.9 | 0.010 | 0.9 | 0.3, 1.5 | 0.002 |

Adjusted for age and body mass index

to 67 controls without clinical cardiovascular disease. We recently assessed  $\underline{112}$  post-menopausal women with PAH age- and body mass index-matched to 148 controls. DHEA-S levels were significantly (50%) lower in PAH cases vs. controls in both men (p = 0.001) and women (p < 0.0001) (Figure 4). Similar to our published findings in men, every 10 Ln( $\mu$ g/dL) decrease in DHEA-S levels increased the odds of PAH by 26% (95% confidence interval 13%–39%, p < 0.0001) in women.

In both men and women, lower levels of DHEA-S were associated with more severe disease including markers of RV function (Table 3). For example, each 1  $Ln(\mu g/dL)$  decrease in DHEA-S levels was associated with a 3 mm Hg higher RAP (p = 0.020) and a 3 Wood unit higher PVR (p = 0.010) in men, and a 2 mm Hg higher RAP (p = 0.019) and 1 Wood unit higher PVR (p = 0.002) in women. The



relationships between DHEA-S levels and markers of disease severity were more robust in women than in men. In women, each 1 Ln ( $\mu$ g/dL) decrease was associated with a 30 meter shorter 6MWD (p = 0.013) (approaching the minimal clinically important difference in PAH)<sup>102</sup>, as well as a 4 mm Hg increase in mPAP (p = <0.001), and may have been associated with a 0.2 L/min decrease in cardiac output (p = 0.067), a trend that was also noted in men. There was also a borderline significant inverse relationship between levels of DHEA-S and functional class in women (Figure 5); patients with lower DHEA-S levels had more symptoms (higher functional class).

It was possible that DHEA-S was exerting effects via E2. However, there was no significant correlation between DHEA-S levels and E2 levels in men (r = -0.15) or women (r = 0.05) with PAH (Figure 6). In addition, the associations between DHEA-S levels and the risk of PAH and all clinical severity measures were unaffected when E2 was added to the models, indicating the demonstrated

Figure 6. Lack of correlation between DHEA-S levels and estradiol levels in men and women with PAH.

Women r = -0.15, p = 0.49

Women r = 0.05, p = 0.43

Ln(DHEA-S), µg/dL

relationships were independent of E2 (and other hormones). There were also no significant interactions between DHEA-S levels and E2 levels (and other hormones) and the risk of PAH nor disease severity markers. In other words, E2 levels did not modify (or mediate) the relationships between DHEA-S levels and PAH risk or disease severity. Lower levels of DHEA-S may contribute to RV remodeling and fibrosis, with downregulation of NO and enhanced ET-1, explaining why lower levels DHEA-S are linked to overall PAH risk and greater severity of PAH and RV dysfunction leading to reduced 6MWD and worse functional class. These data establish a very strong scientific premise in both men and women to treat PAH patients with DHEA to improve clinical outcomes.

**C4. Sex hormone manipulation in human PAH.** In a small (n = 18) study, we have shown that the aromatase inhibitor anastrozole lowered E2 but had no effect on RV function (measured by echocardiographic parameters and BNP) and increased 6MWD.<sup>15</sup> Anastrozole reduced E2 but had no effect on circulating levels of DHEA-S (which may directly impact on NO, ET-1, the pulmonary vasculature and the RV); levels of DHEA-S and E2 are not related and DHEA-S had a direct effect on PAH risk and disease severity wholly independent of E2 levels. A larger, longer Phase II trial of anastrozole in PAH is planned (R01 HL134905; PI Kawut). While our pilot anastrozole study demonstrates the feasibility of sex hormone manipulation as a treatment strategy in PAH, there is no overlap in scientific premise or hypothesized mode of action for DHEA. For these reasons, studies of E2 blockade are complementary to our aims but do not address the therapeutic or mechanistic potential of DHEA in PAH.

C5. Feasibility of collection and characterization of PAECs. Last, we sought to develop mechanistic experiments to explore sex-based differences in patients with PAH. We enrolled patients undergoing right heart catheterization for clinical purposes to isolate PAECs from pulmonary artery catheter (PAC) tips. 103 We first confirmed the presence of non-erythroid cells with counts varying from 25K–968K. We



next confirmed PAEC phenotype (CD146<sup>+</sup>/CD31<sup>+</sup>/CD45<sup>-</sup> and acetylated low density lipoprotein [AcLDL] uptake, von Willebrand factor [vWF] and vascular endothelial-cadherin [VE-cad] staining) in additional samples (Figures 7-8). The NO Metabolomics core (University of Pittsburgh; collaborator Shiva) measured nitrite and nitrate levels in cells with confirmed PAEC phenotype (CD146<sup>+</sup>/CD31<sup>+</sup>/CD45<sup>-</sup> cells sorted; 8K cells) from culture media

with excellent reproducibility (Table 4). Levels were consistent with those that mediate cellular signaling and suggest active secretion of NO.<sup>104, 105</sup> In our most recent experiments, we have isolated ~5 million cells in 3-4 passages and PAECs have remained viable up to 28 days (Figure 8C).

**C6. Summary.** The above studies are among the first to correlate sex and sex hormones (particularly DHEA) to pulmonary vascular and RV phenotype differences in men and women in both health and PAH. This proposal seeks to leverage a safe and available hormone treatment to gain further insight into 4) DV effects (a payel and printiple) and point in DI and DV

**Figure 8.** A. Phase microscopy image, 1 week in culture. B. AcLDL uptake of confluent cells, 2 weeks in culture. C. vWF (green), and VE-cad (red) staining, 4 weeks in culture (20x).



Table 4. NO metabolite levels

| Sample | Nitrite, µM | Nitrate, µM |
|--------|-------------|-------------|
| 1 | 0.27 | 4.95 |
| 2 | 0.26 | 4.99 |
| 3 | 0.27 | 4.97 |
| 4 | 0.25 | 4.83 |
| CV | <1% | <1% |

CV=coefficient of variation; n=500 cells/sample

further insight into 1) RV effects (a novel and critical end point in PH and PAH), 2) effects on two key PAH pathways *in vivo* and *in vitro* as a means for understanding sex-based differences in PAH, and 3) efficiency planning for a future Phase II parallel trial of DHEA as a novel treatment strategy in PAH.

**C7. Investigative team.** The team assembled has expertise in clinical and translational research in PAH and RV failure. This group has collaborated for over five years in the areas of sex hormones, endothelial cell and vesicle biology, and cardiopulmonary function with funding and publications in these areas as well as participation in PAH clinical trials.<sup>5, 101, 106-109</sup> Collaboration with the NO Metabolomics core at Pittsburgh will greatly enhance measurement of NO end points in human and PAEC samples.

#### **C8.** Experimental Plan

**C8.a.** Study design. We propose a "proof-of-concept" crossover study to examine the safety and efficacy of 50 mg daily of DHEA for 18 weeks in patients with World Health Organization (WHO) Group

1 PAH (Figure 9). The primary outcome is RV longitudinal strain. Secondary outcomes include the effects of DHEA on markers of RV remodeling (**Aim 1**) as well as HRQOL, other PAH end points, side effects and safety. We will determine DHEA's effects *in vivo* in the cross-over trial (**Aim 2**) and *in vitro* on NO and ET-1 pathways in PAECs from subjects with PAH and whether these effects differ by sex (**Aim 3**)

C8.b. Scientific rigor. The selection of the cross-over design by definition eliminates between-subject variability when comparing drug to placebo and allows for a much smaller sample size than would ordinarily be necessary (e.g., in a parallel arm trial) to maintain the same power. Since each subject acts as their own control, it also prevents against the imbalance of



other important factors related to rigor, namely age and race/ethnicity. However, differences in drug effectiveness by age, sex, etc. can still be assessed. This design will also allow us to examine patient-level responses in carefully selected end points (imaging, biomarker, functional, HRQOL) so that we may assess for potential interactions by age and race/ethnicity (as well as sex and PAH sub-type) and time by treatment effects while reducing variability and improving precision.

Study end points are subject to measurement error and missingness. Measurement error will be minimized by using validated methods with demonstrated precision in experienced laboratory and imaging cores with QC in place. Every effort will be made to minimize missing data via study procedures, close follow-up, and subject retention efforts. Bias will be minimized by masking patients, investigators, and personal and randomizing the treatment periods. While the proposed sample size is small, the cross-over design by definition optimizes statistical efficiency and minimizes confounding given each participant is their own control and treatment order is randomized. Multiple comparisons could result in Type I error, but our power calculations are based on distinct hypotheses about RV phenotype. Because of the cross-over design, small differences are likely to be detected making Type II error unlikely.

**C8.c.** Subjects. We will randomize 26 subjects stratified by sex (13 women, 13 men) and PAH type (idiopathic PAH vs. other) from the Rhode Island Hospital Pulmonary Hypertension Center (RIHPHC) to active treatment

(Period 1), placebo (Period 2) or to placebo (Period 1), active treatment (Period 2) (Aims 1, 2). PAH patients meeting the same inclusion criteria (Table 5) undergoing hemodynamics will be eligible for PAEC collection (Aim 3).

C8.d. Inclusion/Exclusion criteria (**Table 5**). Patients on PAH therapy will be enrolled provided they have had no new PAH therapies introduced for 12 weeks (see Table 5 for specifics). We will include premenopausal women but will track menstrual cycle dates and measure sex hormones at each visit; physiologic variations should be balanced by the cross-over design (i.e., at least four to five menstrual cycles per 18 week treatment assignment). At least four weeks of clinical stability (no hospitalizations or titration of PAH therapies) will be required prior to randomization. Additional exclusion criteria speak to the elimination of other types of PH (#2, 5-6) or conditions in which DHEA is untested (#7-8) or has uncertain or potentially harmful effects (#1, 9-11). Indwelling (>3 months) levonorgestrel IUDs will be allowed. The progestin effect of hormonereleasing IUDs occurs primarily at the endometrium<sup>147</sup>. Serum hormone levels can be affected transiently (out to seven days postinsertion) but there is gradual decline over time which stabilizes. In a potential female subject with a long-term (3 months-5 years) hormone-containing IUD in place, systemic progestin levels are stable and, especially given the cross-over design, should not confound results.

#### Table 5. Inclusion and Exclusion Criteria

#### Inclusion Criteria

- mPAP ≥ 25 mmHg at rest, pulmonary capillary wedge pressure or left ventricular end-diastolic pressure ≤ 15 mmHg, and PVR > 3 Wood units at any time prior to study entry.
- Diagnosis of PAH that is 1) idiopathic, 2) heritable or 3) associated with connective tissue disease, congenital systemic-to-pulmonary shunt, portopulmonary hypertension, drug or toxin use
- Pulmonary function testing documenting forced expiratory volume in one second/forced vital capacity ratio ≥ 70% predicted, total lung capacity ≥ 70% predicted.
  - If TLC is mildly reduced (60%<TLC%<70%), computerized tomography (HRCT or non-HRCT) documenting no significant interstitial lung disease may be used to fulfill this requirement.
- Chest tomography documenting no more than moderate parenchymal lung disease with clinician designated WHO I PAH and meeting both TLC and FEV1/FVC criteria.
- Ventilation/perfusion (V/Q) testing documenting absence of thromboembolic disease (normal or low probability V/Q scan)
  - If no V/Q scan is available, a CT angiogram documenting the absence thromboembolic disease may be used, provided the subject meets diagnostic PAH criteria (as above).

#### **Exclusion Criteria**

- 1. Age < 18 years old
- 2. PAH associated with human immunodeficiency virus infection
- 3. Initiation of new background PAH therapy within 12 weeks of baseline visit
- 4. Significant dose change in background PAH therapy. The following ARE allowed:
  - a. within 12 weeks of baseline visit:s
    - i. planned titration of prostacyclin analogue, selexipag, or riociguat >20%
    - ii. Plan to titrate to high dose sildenafil (e.g., 20mg to 80mg TID)
    - iii. Transition to prostacyclin analogues/selexipag (e.g., IV to oral, inhaled to IV)
    - iv. Increase in ambrisentan 5mg to 10mg or tadalafil 20mg to 40mg
  - b. within 4 weeks of baseline visit:
    - i. planned titration of prostacyclin analogue, selexipag, or riociguat <20%
    - ii. change from commercial to generic (or generic to commercial) ERA or PDE5i iii. Interchange within drug class due to side effects (e.g., ERA to ERA, PE5i to
  - iii. Interchange within drug class due to side effects (e.g., ERA to ERA, PE5i t PDE5i)
- 5. Untreated severe obstructive sleep apnea diagnosed by polysomnography
- Evidence of left-sided valvular disease or systolic dysfunction on echocardiogram (≥ moderate mitral or aortic disease or LV ejection fraction ≤ 50%)
- 7. Glomerular filtration rate <40 mls/min/1.73m<sup>2</sup>
- 8. Child-Pugh Class C cirrhosis
- 9. Untreated hypo- or hyper-thyroidism
- 10. Pregnant or breastfeeding
- 11. Active or planned use of hormonally active therapies with the exception of indwelling (>3months) levonorgestrel IUDs (see Appendix A for list of excluded medications and hormonal therapies).
- 12. History of breast, ovarian, uterine, testicular or prostate cancer
- 13. Current use of another investigational PAH therapy
- 14. Contraindication to MRI (e.g. metal device or fragment)
- 15. History of significant non-adherence or circumstance which would threaten ability to comply with cross-over design and study visit schedule

**C8.e.** Subject recruitment and retention. The RIHPHC services a catchment area of all of Southern New England and is the only center accredited by the Pulmonary Hypertension Association as a Comprehensive Care Center in the region. The RIHPHC cares for >400 patients and offers comprehensive patient care services including diagnostic imaging, hemodynamic evaluation, a dedicated PH step-down unit, an interdisciplinary care team, and four full-time providers. The PI and staff of RIHPHC meet weekly to screen patients for enrollment in active research protocols. Eligible patients will be approached by their PAH clinician and then by the PI or research staff. Following screening and informed consent, a maximum of four weeks may lapse before randomization (baseline visit) and eligibility in order to confirm clinical stability. New or recent changes to PAH meds will be reassessed at the baseline visit. Serum pregnancy tests will be obtained at

baseline and at week 24 (after crossover) in premenopausal subjects. Retention and complete follow-up will be assured with frequent call reminders 3-5 days prior to study visits, 24/7 accessibility of research support staff, study drug adherence logs and pill counts, and monetary compensation and parking passes for study visits.

PAH in men is rare, however based on our trial enrollment over the past three years (n = 52, 25% men) and our recent study of men<sup>101</sup> we anticipate recruiting 13 (50%) men during the study. Patient-level variation in end points as well as interactions by age, sex, race/ethnicity, and PAH sub-type will be assessed. We have met all of our enrollment targets for active studies, and consider this proposal a top priority for our center.

**C8.f.** Investigational therapy. We have already received an Investigational New Drug exemption (IND#129285) from the FDA for this study (see attached letter). We will purchase DHEA 50 mg daily tablets in a single batch from Green Mountain Pharmaceuticals (Lakewood, CO), Green Mountain is an Active Pharmaceutical Ingredient registered manufacturer with the FDA and has produced DHEA for ongoing trials at major centers including our institution (NCT01343771). Lots previously purchased

| Table 6. Study protocol and | end points | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Timeline, week | | 2 | 18 | 19-22 | 24 | 40 | 42 | Unscheduled |
| Study visit | Baseline | #1 | #2 | Washout | #3 | #4 | | US |
| Phone call | | | Χ | Х | | | Х | |
| Medical history | X | | | | | | | |
| Medications | Х | Χ | Χ | | Χ | Χ | | X |
| History and physical exam | X | Χ | Χ | | Х | Χ | | X |
| Laboratory/safety | | | | | | | | |
| CBC, Chem 7, hepatic | X | Χ | Χ | | Χ | Χ | | as indicated |
| Hormone levels | X | Χ | Χ | | Χ | Χ | | as indicated |
| Insulin levels | X | Χ | Χ | | Χ | Χ | | as indicated |
| Cholesterol levels | X | Χ | Χ | | Χ | Χ | | as indicated |
| Triglyceride levels | X | Χ | Χ | | Χ | Χ | | as indicated |
| End points | | | | | | | | |
| Aim 1: Cardiac MRI | X | | Χ | | | Χ | | |
| Aim 1: NT-proBNP,<br>galectin-3, RAGE, redox | X | X | Х | | Х | X | | |
| Secondary: SF-36v2,<br>emPHasis-10, FC, 6MWD | X | Х | Х | | Х | Х | | |
| Aim 2: NO-related markers | Х | Χ | Χ | | Χ | Χ | | |
| Aim 2: ET-1 | Х | Χ | Χ | | Χ | Χ | | |
| Study procedures | | | | | | | | |
| Dispense study drug | Х | | | | | | | |
| Medication adherence | | Х | Х | | Χ | Χ | | |

from this manufacturer yielded >100% DHEA from an independent laboratory (FrontRangeLabs, Loveland, CO) (included with IND letter). We will also analyze and document purity in the batch purchased for this study. Study drug and placebo will be over-encapsulated by the Investigational Services Pharmacy (see letter of support). Dose, 18 week exposure and four week washout periods were chosen based on pharmacokinetics of DHEA, treatment duration required for RV changes, and early phase trial standards in endocrine and PAH. 10-113 Changes in RV function occur after just 12 weeks of PAH therapy, justifying the planned exposure period. 36

Adverse events

**C8.g. Study protocol and burden.** An 18 week supply of study drug will be dispensed following randomization at the baseline visit. Cardiac MRI for RV measures (Aim 1) will be assessed at baseline, week 18 and week 40, at the end of each period receiving active treatment or placebo. Laboratory (Aim1: NT-proBNP, galectin-3, RAGE, oxidative stress markers and those for safety; Aim 2: plasma NO-related markers and serum ET-1) and secondary end points will be assessed at baseline and all four study visits (Table 6). Data collection for history and physical exam, adherence, and adverse events will occur in the RIHPHC research room, followed by 6MWD in the RIHPHC hallway. Phlebotomy for study labs will be performed by trained personnel and cardiac MRI will be performed at the end of the visit in the MRI suite; labs and imaging will occur on the first floor of the same building where the RIHPHC is located. Subjects will complete the HRQOL measures on a tablet during downtime to r educe total visit time. We will offer a small meal after phlebotomy. Based on current protocols including similar tests we anticipate the total time for a study visit will be 90–120 min (visit #1, #3) and 210–240 min for visits with MRI (baseline, visit #2, #4).

**C8.h. Drug and protocol adherence.** Pill counts will be tracked at each visit. A phone call after visit #2 at week 18 will confirm plan for the washout period. A second call in the washout period prior to visit #3 will ensure start date for second course of study drug.

**C8.i.** Randomization and blinding. Randomization of drug sequence stratified by sex and PAH subtype (Period 1–Period 2; Period 2–Period 1) will be automated by a web-based program. Study personnel and

subjects will be blinded to treatment order allocation. DHEA and placebo will have identical packaging, taste. and smell. Study drug will be dispensed at the start of each treatment phase (weeks 0-18 [Period 1]; 22-40 [Period 2]) with phone calls as outlined.

- C8.j. Safety monitoring. The research coordinator (Amy Palmisciano RN, BSN) and research assistant will be available 24/7 by phone as needed for side effects and adverse events. An unscheduled study visit can also be performed if lab abnormalities on safety labs require retesting. Provisions for an unscheduled study visit can be found in Table 6. RIHPHC clinicians and research staff including the study PI will be capable of breaking the blind in case of an adverse event. A data safety monitoring board (DSMB) consisting of three independent clinician scientists with expertise in cardiology, pulmonology and/or endocrinology and a biostatistician with clinical trial experience will be assembled to review enrollment targets, protocol deviations, violations, and adverse events as described below. Conference calls will occur throughout the study period and on an as needed basis for serious adverse events. Please see Section C8.m.6. for specific safety end points and Data and Safety Monitoring document for further details.
- C8.k. Drop-out. Subjects may end participation by completion of the trial, loss-to-follow-up, withdrawal of consent, or death. In the last three RCTs conducted at our center (n = 21) we have had no patients lost to follow-up (rare in this patient population) and two patients (11%) withdraw. In our power calculations, we have anticipated a 10% drop-out rate; any subjects who need to withdraw from the study will continue study assessments whenever possible and be analyzed in an intent-to-treat fashion.
- C8.I. Outcomes for the crossover trial. The primary outcome will be changes in longitudinal strain with DHEA (Aim 1). Secondary outcomes will include RVEF, NT-proBNP, galectin-3, RAGE, MPO and sNOX2-dp levels (Aim 1), sex hormone levels, HRQOL, WHO functional class, 6MWD, side effects, and safety of DHEA in PAH. We considered using right heart catheterization as a study end point but given the cross-over design (which has benefits in terms of power and precision) this would require three right heart catheterizations which poses undue burden on (and risk to) participants and a threat to feasibility. Additional end points (e.g., HRQOL) were selected based on prior DHEA trials demonstrating efficacy in similar disease states with high relevance to PAH. Aim 2 outcomes will include changes in NO and ET-1 molecules with DHEA treatment.
- C8.I1. Aim 1: Longitudinal strain and RVEF. We have a core MRI facility with a Siemens 1.5T Aera with full Advanced Cardiac Package and XJ Gradients (33 mT/m @ 125 T/m/s) that provides research grade studies at a greatly reduced cost. A single reader (Michael Atalay, MD, PhD) will be blinded to subject and study visits and will read studies in randomly sequenced batches; 10% of the studies will be re-read by the same reader and 10% of scans will be re-read by a second reader for intra-reader and inter-reader reliability estimates. Dr. Atalay's research focuses on cardiac MRI and he is experienced in RV imaging in PAH. A standardized MRI protocol is proposed:
- 1) Quantification of end-diastolic volume (EDV), end-systolic volume (ESV), EF, and mass. Shortaxis steady state free precession from the base of the heart through the apex (Figure 10). All analyses will be performed using commercially available cardiac MRI software (CVI42, Circle Cardiovascular Imaging). The endocardial and epicardial borders of both ventricles will be traced manually on short axis cine images at end-diastole and end-systole. EDV and ESV will be calculated using Simpson's rule by summation of areas on each slice multiplied by the sum of slice thickness and image gap. Ventricular EFs will be calculated by dividing respective stroke volumes (EDV-ESV) by EDVs. RV and LV mass will be determined at the end-diastole phase as the

difference between end-diastolic epicardial and endocardial volumes X heart specific gravity  $(1.05 \text{ g/cm}^3).^{114}$ 

2) Quantification of pulmonary insufficiency, independent quantification of RV stroke volume and measurement of main PA cross-section through the cardiac cycle (distensibility). Breath-hold through-plane phase contrast imaging with a velocity encoding gradient (VENC) of <120 cm/s (larger if aliasing



Figure 10. Short axis cine images for







Figure 11. Through-plane phase contrast for main PA distensibility

present) in the main PA ~2-3 cm above the pulmonary valve plane, with imaging plane oriented orthogonal to the main PA (Figure 11). Free-breathing phase contrast imaging in the same plane and VENC with averaging over 4 respiratory cycles.

**3)** Longitudinal and circumferential strain will be determined using standard cine imaging and MTT software (version 6.0, Toshiba, Japan). This program utilizes a pixel-matching algorithm to define angle-independent motion vectors from multiple tracking points for location of identical voxels in serial frames (Figure 3). Algorithm will be repeated twice for each subject and include biventricular borders throughout the cardiac cycle. Peak systolic segmental strain will be extracted from inner, mid, and outer walls. **C8.12. Aim 1: Markers of RV Phenotype.** Blood via venipuncture will be collected by trained staff. Samples will be processed and stored at -80°C. Serum NT-proBNP levels will be measured using a FDA approved commercially available immunoassay (Roche Diagnostic Elecsys proBNP Assay, Indianapolis, IN) with excellent precision (intra- and inter-assay CV of <6.1%) and a track record in PAH.<sup>115, 116</sup> Serum galectin-3 levels will be measured by an enzyme linked immunoassay (ELISA) with an intra-assay CV of 3.4% (BG Medicine, Waltham, MA). Soluble RAGE levels in plasma will be measured by an ELISA (R&D Systems, Minneapolis, MN) with excellent precision (intra-assay CVs 4.8% – 6.2%; inter-assay CVs 6.7% – 8.2%). Serum MPO levels will be measured by a commercially available ELISA (CardioMPO Test, Prognostix, Cleveland, Ohio) and sNOX2-dp by ELISA using previously published methods, both with excellent precision.<sup>72</sup>

#### C8.m. Secondary outcomes for the crossover trial

**C8.m1. HRQOL.** Patient-reported outcomes as assessed by HRQOL measures provide important information not captured by traditional surrogates and especially relevant in PAH, a progressive disease without cure treated with burdensome and side effect-laden therapies. The **SF-36v2** is a widely used instrument that provides information about HRQOL along 8 domains condensed into physical and mental component summary scores. The SF-36 and its updated version SF-36v2 has been validated in chronic diseases including PAH, has been used as a secondary end point in RCTs of approved PAH therapies, and tracks with survival. <sup>117-123</sup> **emPHasis-10** is a PAH-specific HRQOL tool that is uni-dimensional and pragmatic (10 items). It is sensitive to clinical changes in PAH and has been translated into multiple languages with cultural and linguistic validation. <sup>124, 125</sup> Subjects will be asked to complete the SF-36v2 and the emPHasis-10 at each research visit (Table 6). Changes from baseline in domain-specific scores and summary scores for the physical and mental components for the SF-36v2 and the summary score for emPHasis-10 will be assessed.

**C8.m2. WHO Functional class.** Functional classification drives initial choice of therapy and is a major treatment goal in PAH. <sup>126</sup> WHO class is derived from the New York Heart Association classification: Class I is no limitations; Class II is slight limitations in physical activity and no symptoms at rest; Class III is symptoms with minimal activity; Class IV is symptoms at rest. Clinicians will assess functional class at each study visit.

**C8.m3. 6MWD.** Change in 6MWD has been the primary end point for almost all Phase III trials and the basis for drug approval in PAH.  $^{127}$  Testing will be performed by blinded and trained personnel according to standardized procedures.  $^{128}$  We will minimize variability by administering the test in the same corridor for all subjects, avoiding a "warm-up" period, and using standard phrases of encouragement; intra-class correlation coefficients were 0.95-0.98 from a recently completed RCT in our center (NCT01545336).

**C8.m4. Sex hormone levels.** We will measure serum sex hormone levels at baseline and with each study visit to capture overall changes in the hormonal mileau during active treatment and placebo phases using highly sensitive assays with excellent QC as we have previously reported.<sup>15, 101</sup> DHEA-S (more stable than DHEA in biosamples) will be measured on the Immulite 2000 analyzer (Siemens Healthcare Diagnostics, Deerfield IL).

**C8.m5.** Additional signaling molecules of interest. Given experimental PH models have linked DHEA to important signaling pathways in the immune and fibroproliferative components of PAH (e.g., IL-6, MAPK, STAT3), we will investigate whether DHEA treatment impacts serum IL-6 and soluble IL-6 receptor levels using commercial ELISAs. <sup>19, 20, 65, 129</sup> PAEC experiments will also assess MAPK and STAT3 signaling (Section C9.).

**C8.m6.** Side effects and safety. Study personnel will assess side effects and adverse events by body system during each visit and in phone calls during the washout phase and end of study call at week 42. We will specifically query participants about potential known side effects of DHEA, such as androgenic symptoms (change in skin/greasy skin, acne, alopecia and/or hirsutism) and we also assess HRQOL from these potential side effects as outlined above with the SF-36v2. Laboratories to assess for safety will include: complete blood count, complete metabolic panel, glucose levels, insulin levels, liver function tests, high density lipoprotein, low

density lipoprotein, total cholesterol and triglyceride levels using standardized assays. While we do not anticipate drug-related adverse events, in all cases the referring and/or primary care physician will be notified in writing of the adverse events, the subject's status, and receive a copy of laboratory abnormalities, as appropriate. Study drug will be continued for mild side effects such as androgenic symptoms. A detailed monitoring plan will be submitted to the local IRB before the trial begins in accordance with NIH/NHLBS policy for early phase trials and will include mechanisms for adverse event reporting to the IRB, the FDA, and the NIH (see Human Subjects Protection). No interim analysis is planned for this pilot study.

C8.m7. Aim 2: NO-related molecules. NO synthesis will be assessed by the NO Metabolomics core facility (University of Pittsburgh; collaborator Shiva). Plasma nitrite and nitrate levels will be quantified using tri-iodide-based reductive chemiluminescence. 105, 130, 131 Whole blood will be immediately processed with a readily available precooled centrifuge to 4°C after the addition of nitrite preservation. 130 Care will be taken to avoid sample exposure to light and to use nitrite-free equipment. The specific contribution of nitrite will be calculated by subtracting nitrosocompounds from the total chemiluminescence signal after treatment with acidic sulfanilamide. We additionally propose to measure interrelated molecules in the NO pathway known to be abnormal in PAH including cGMP levels and S-nitrosohemoglobin (SNO-Hb), a major regulator of NO's interaction with vascular endothelium. 132-135 cGMP will be measured via immunoassay (Biomedical Technologies, Inc, Madrid, Spain). 136 SNO-Hb levels will be measured using chemiluminescence as for nitrites and nitrates; these methods have been well-validated by the NO Metabolomics core facility. 131

A <u>potential pitfall</u> is that the direct measurement of steady state NO is difficult due to endothelial and cellular metabolic flux and rapid half-life. As such the sum of nitrates and nitrites are not necessarily reflective of total NO synthesis activity and may capture changes in diet or external contamination, for example. <sup>137</sup> The measurement of nitrates is subject to such interference, whereas as much as 90% of circulating nitrites in plasma is the result of the L-arginine-NO production pathway. The NO Metabolomics core facility at the University of Pittsburg has extensive experience in assessing pulmonary vascular NO and employs state-of-the art approaches to ensure accuracy and precision known to be <u>more sensitive for NOS signaling than other methods (especially from banked samples) including electron paramagnetic resonance. <sup>130, 138</sup></u>

**C8.m8. Aim 2: ET-1.** Serum ET-1 will be measured via immunoassay (QuanitGlo, R&D Systems, Inc, Minneaopolis, Minn) with intra-assay CVs of 2.6 - 3.4% and inter-assay CVs of 4.6 - 8.9%.

- **C8.n. Data collection and management.** Our clinical research coordinator will oversee data collection and management. She has extensive experience working in pulmonary/critical care clinical-translational research and specifically in PAH for the past four years. All data will be collected in a secured fashion with paper case report forms and immediately transposed to an electronic system (REDCap) to ensure back-up. Data will be stored on a secure server. Plan for data sharing with the University of Pittsburgh is described in the Plan for Resource and Data Sharing and Human Subjects Protection documents. The PI will be responsible for data security and cleaning; analysis will be completed by G. Baird, PhD who has collaborated closely with the PI.
- **C8.o.** Analysis plan for the crossover trial. Demographics and clinical data will be provided, stratified by sex as well as PAH subtype. This data will also be tracked for screen failures and drop-outs. Continuous data will be expressed as medians and ranges and categorical data will be expressed as frequency and percentages. Analyses will follow the intention-to-treat paradigm. All end points will be modeled using generalized estimating equations (GEEs), nesting repeated measures within patient and including terms for sex, age, race/ethnicity, PAH-subtype, randomization, and time point, along with all 2-way and 3-way interactions in which carry-over or period effects will be considered. Distribution will be chosen based on inspection of model residuals. Classical sandwich estimation will be used to adjust for model misspecification after maximizing the appropriateness of distribution selected. Orthogonal linear estimates will be constructed within GEEs to test each hypothesis (see Aims) and presented both as the percentage change and absolute change in RV measures (Aim 1), changes in NO products and ET-1 (Aim 2), and secondary end points. No adjustment for multiple comparisons will be made given the pilot nature of the study. The main effect of DHEA and interactions of DHEA with sex (as well as age, race/ethnicity, PAH-subtype) will be tested within models, with use of visualizations including individual scores for exploratory analysis. Hypotheses will be two-tailed.
- **C8.p. Sample size and power for the crossover trial.** We anticipate a 10% drop-out rate and calculated power based on an anticipated sample size of 24 subjects (12 men, 12 women). As this is a pilot study, detection of a signal (even if not statistically significant) and "proof of concept" that DHEA treatment may improve RV phenotype and alter major PAH regulators would encourage the pursuit of a

larger Phase II parallel arm trial. Time by treatment and PAH subtype by treatment interactions will also be

considered as part of 3-way interactions terms in GEE.

Table 7. Power calculations for RV strain (N = 24)

| | | RV strain difference, % | Power |
|---|---|---|---|
| C8.p1. Aim 1: Power to detect differences in RV longitudinal | No | 3.0 | 89% |
| <b>strain.</b> We will have excellent power to detect clinically relevant | interaction | 5.0 | 99% |
| changes in RV strain ( $\alpha = 0.05$ )(Table 7). A $\geq 5\%$ improvement | | 7.0 | 100% |
| in RV strain (measured by echocardiography; less precise than | Interaction | 4.0 | 80% |
| MRI) occurs with approved PAH therapies and predicts clinical | | 5.0 | 94% |
| stabilization and survival in PAH. <sup>56</sup> We have more than enough | | 7.0 | 100% |
| Stabilization and deriver in 1741. We have more than energy | | | |

power to detect this estimate, and effects even as small as 3%. We need this number of patients in order to perform sex-specific analyses (and test for treatment x sex interaction), where we will have 80% power to detect a 4% difference in sex-specific analyses

 Table 8. Power calculations for RVEF and NT-proBNP (N = 24)

| | RVEF, % | Power | NT-proBNP, mg/L | Power |
|----------------|---------|-------|-----------------|-------|
| No interaction | 5.0 | 80% | 200 | 98% |
| Interaction | 8.0 | 80% | 200 | 80% |

with the presence of an interaction. Power for treatment x PAH subtype interactions will mirror these estimates. We will also have sufficient power to detect changes which approach clinical relevance in RVEF<sup>61, 139</sup> and NT-proBNP<sup>140</sup> ( $\alpha = 0.05$ ) (Table 8).

C8.p2. Aim 2: Power to detect differences in nitrate and ET-1 levels. We will have excellent power to detect small (0.05  $\mu$ M) differences in nitrite levels with DHEA treatment based on conservative previously observed estimates ( $\alpha$  = 0.05).<sup>25, 141</sup> We will have excellent power to detect small (well-less than 2 pg/mL) differences in ET-1 levels with DHEA treatment ( $\alpha$  = 0.05). Changes of this magnitude would be consistent with clinically relevant changes in ET-1 with ERAs.<sup>142</sup>

C9. Aim 3: PAEC response to DHEA. In order to minimize burden of the trial participants (and to guarantee more catheter tips), PAECs from men and women undergoing right heart catheterization at the RIHPHC as part of PAH diagnosis or treatment and meeting the same inclusion/exclusion criteria for the cross over trial will be included. As with our preliminary data, these experiments will be performed in our Centers of Biomedical Research Excellence in Stem Cell Biology (PI: Quesenberry, P20 GM103468) and



Cardiopulmonary Vascular Biology (PI: Rounds; Laboratory Core PI: Harrington, P20 GM103652). We will also examine the effect of DHEA on PAECs obtained from two additional sources: 1) commercially available human PAECs, 2) those obtained from the distal pulmonary circulation of PAH lung explants available through the Pulmonary Hypertension Breakthrough Initiative (PHBI) (PI Geraci, R24 HL123767; see letter of support).

We will isolate PAECs and assess NO and ET-1 production at baseline and following exposure to DHEA (Figure 12). Following catheterization, the PAC tip will be placed into 1 well of a 24 well plate, with Attachment Factor Solution (Cell Applications, Inc, San Diego, CA) and media (EndoGRO, Millipore Sigma, Billerica, MA). The PAC tip will be washed with fresh media every 2 days and previous media from the tip well will be moved into a new well in the 24 well plate. Cells will be grown in primary culture to confluence (~150K-200K cells) over 2-3 weeks. Cells will then be treated with Triple Express (ThermoFisher Scientific, Waltham, MA) and transferred to T-25 and then T-75 flasks over 4-5 days; we anticipate ~5 million cells in 3-4 passages. In the event that we are unable to culture a robust number of PAECs using the above protocol, conditioned media charcoal-stripped of all steroid hormones will be used.

- 1) NO and ET-1 synthesis. Cell lysate and culture media from cultured PAECs passage 3-5 will be snap frozen in liquid nitrogen and stored at -80°C. ET-1 and cGMP will be measured by ELISA and nitrite and nitrate levels will be quantified using tri-iodide-based reductive chemiluminescence (See Section C8.m7). Expression of eNOS, soluble guanylyl cyclase (sGC)  $\alpha$  and  $\beta$ , IL-6, STAT3, and MAPK will be measured with standard RT-PCR and Western blot methods using commercial nucleic acid probes and antibodies.<sup>144</sup>
- **2) Cell treatment.** Cells will be incubated at  $37^{\circ}$ C in media in the presence or absence (controls cells) of DHEA at final concentrations of 1, 10, and 100  $\mu$ M (Sigma-Aldrich, St. Louis, MO). Initial experiments will be conducted using commercially available PAECs to determine optimum cell concentration and exposure times that will provide consistent assessment of NO and ET-1 synthesis. Cell proliferation, migration, adhesion, and tube formation will be characterized before and after exposure to DHEA using standardized protocols

performed in our laboratory<sup>145</sup> with concurrent confirmation of PAEC phenotype. We will also determine the effect of DHEA in commercially available disease free PAECs. These conditions will then be used in experiments to assess DHEA's effects on NO and ET-1 synthesis in PAECs from both sexes with PAH. All experiments will be repeated with 1) exposure to E2 for comparison and 2) in PAECs from lung explants to determine if distal and proximal PAECs respond in a similar way to DHEA.

**C9.a. Analysis Plan Aim 3: PAEC response to DHEA.** Wilcoxon signed-rank tests and analysis of variance will be used to compare ET-1 and eNOS expression and nitrite and nitrate levels before and after DHEA treatment and across cells from men and women.

**C10. Study timeline.** Based on prior recruitment rates and fractions, we will be able to enroll 4-7 subjects per year as outlined in the study timeline. A five year mechanism is proposed and is needed in order to ensure adequate inclusion of men and completion of the protocol for subjects recruited later in the study period to allow adequate time for follow-up, biomarker and data analysis (which cannot be completed until all subjects enrolled later in the study complete the 42 week crossover trial protocol).

C11. Expected results
C11.a. Aims 1 and 2. Active
treatment with DHEA will be
associated with an improvement
in RV strain pattern, lower ET-1
levels and higher nitrite and nitrate
levels. Markers of maladaptive RV
hypertrophy including oxidative
stress will also be reduced. Sex

Table 9. Study timeline

| | Yr 1 | Yr 2 | Yr 3 | Yr 4 | Yr 5 |
|---|---|---|---|---|---|
| Start-up: Drug purity testing | Mos 1-6 | | | | |
| Relational trial database buildout | Mos 1-6 | | | | |
| Policies and Procedures, IRB approval | Mos 1-6 | | | | |
| Aim 1,2: Cross-over enrollment | n = 4 | n = 7 | n = 7 | n = 6 | n = 2 |
| Aim 3: Commercial cells, PHBI | X | Χ | Χ | Χ | |
| Aim 3: PAECs, patient catheterizations | n = 15 | n = 15 | n = 15 | n = 15 | n = 15 |
| Lab/results analysis | | | | Χ | Χ |
| Manuscript/grant preparation | | | | X | Χ |

will modify these relationships, with women demonstrating a more robust response to DHEA.

**C11.b.** Aim 3. NO and cGMP synthesis will be higher and ET-1 secretion will be lower in PAECs from women with PAH than PAECs from men, respectively. Treatment with DHEA will increase eNOS expression and nitrite/nitrate levels and decrease ET-1 secretion. Female cells will demonstrate a more robust and distinct response to DHEA than male cells and E2 exposure respectively.

#### C12. Potential problems and alternative approaches

C12.a. Aims 1 and 2: Clinical trial completion and end point evaluation. Enrollment: A major threat to clinical studies in a rare disease is low enrollment. The RIHPHC has an extensive track record of participation in NIH funded efforts of hormonal modulation in PAH where we have met and surpassed recruitment goals (P20 GM103652 [PI:Ventetuolo] and K24 HL103844 [PI: Kawut; NCT01545336]). 146 We have tried to minimize burden, provided incentives, and prioritized this trial over invitations to participate in others to ensure adequate recruitment. Drop out will be minimized by study procedures and follow-up ensured as PAH patients require highly specialized care available regionally only at the RIHPHC. Study endpoints: In the event that DHEA has no effect on our primary end point, a number of other secondary and exploratory end points have been incorporated which capture alternative markers of interest (e.g., oxidative stress) and will serve to shed light on sexual dimorphism in PAH. We considered measurement of central hemodynamics a lower priority given our interest in studying the direct effects of DHEA on the RV, and felt the burden from repeat right heart catheterizations would threaten feasibility. Intervention: We selected a lower dose of DHEA (50 mg) than given in the prior trial of COPD-PH (200 mg) because the majority of RCTs have used the 50 mg dose with no serious adverse events and minimal side effects. 73, 79 We considered a dose-finding study, but the 50 mg dose has been very well-established as sufficient to increase DHEA-S levels without intolerable side effects. The 50 mg dose has been associated with improvements in biomarkers in atherosclerosis and HRQOL in lupus (as proposed here). A highly pure compound will be verified. It is possible that DHEA may work via alternative mechanisms to those proposed; alternative biomarkers may be tested from banked samples from study visits to be further developed in our cell-based experiments.

**C12.b. Aim 3: PAEC response to DHEA.** This aim will be completed in PAH patients undergoing routine right heart catheterization, which may or may not include patients included in the crossover trial and therefore may

constitute a "missed opportunity" to study results of *in vivo* controlled DHEA exposure *in vitro*. We did not incorporate catheterization into the study protocol in an effort to minimize burden but did restrict eligibility for this aim to match inclusion/exclusion criteria for the trial. We perform dedicated right heart catheterizations in 40 – 60 patients yearly, providing ample opportunities to obtain PAECs from PAH patients. Over the last twelve months since this protocol was initiated, PAEC samples have been collected in 57 patients. The PAECs collected (and their response to DHEA exposure) may not represent the phenotype of PAECs from small resistance vessels in PAH (which will also be included for comparison, Section C9). PAH patients have changes in proximal PAs which contribute to circuit compliance and ventricular coupling<sup>147</sup>, however, making the proposed experiments relevant. Moreover, recent studies using induced pluripotent stem cells from dermal fibroblasts of PAH patients showed that derived endothelial cells function the same as distal PAECs isolated from explanted lungs. PAECs obtained from lung explants represent end-stage PAH, whereas our method captures PAECs from patients at variable stages of disease. Finally, this is a very novel approach with which we have become increasingly facile in a disease state in which tissue availability is extremely limited.

**C13. Summary.** This pilot double-blind cross-over trial will test the efficacy and safety of DHEA in men and women with PAH and will characterize the interaction of sex- and sex-hormones with major pathologic drivers of pulmonary vascular and RV dysfunction. Complementary *in vitro* experiments will offer additional insights into mechanisms of sexual dimorphism in PAH. The first study of its kind, we will build a foundation for sex- and hormone-based treatment precision in this rare and progressive disease.

#### **Amendments and Addendums:**

#### Amendment 1 - PAEC Biobanking and RNA Sequencing

Pulmonary arterial cells (PAECs) collected from catheter tips may undergo RNA sequencing as part of an advanced characterization protocol, representing a continuation of the aims of Aim 3 above. The PAECs for RNA Sequencing will be sourced from the current study's subjects and from a previous biobank (PI: Klinger, IRB Committee #: 016311). Furthermore, all PAEC cultures will be preserved for future, unknown testing and stored in accordance with the Lifespan HRPP Specimen banking guidelines.

#### Amendment 2 – Biobanking for Aim 1 and 2 (clinical trial samples)

A portion of blood collected (in the form of plasma and serum) under Aim 1 and 2 of the protocol ("the DHEA clinical trial") will also be banked. No additional blood will be collected. We will bank the remnant samples after protocol laboratory testing has been performed.

#### Amendment 3 – Unscheduled Visit Provision, Inclusion/Exclusion Clarification and SF-36v2

- 1. Added provisions for an unscheduled study visit in case of clinically significant safety lab abnormalities. Details can be found in Table 6 and section C8.j.
- 2. This amendment also clarifies three inclusion criteria:
  - A. If TLC is mildly reduced (60%<TLC%<70%), computerized tomography can be used in order to rule out any clinically significant interstitial lung disease and allow for inclusion.
  - B. Changes "absence" of parenchymal lung disease to "no more than moderate" disease with the provision that the treating physician has deemed the patient's underlying PAH as unrelated or out of proportion to lung disease (i.e. patient has WHO group 1 PAH) and the patient meets PFT criteria. The PI will verify the validity of all diagnoses.
  - C. If no V/Q scan is available and meets study diagnostic criteria for WHO 1 PAH, a negative CTA Pulmonary Embolism can be used instead.

The above three clarifications put the study in congruence with the diverse phenotypic realities of the PAH patient population. We do not believe these changes will have any impact on the scientific rigor of this study.

All changes are detailed in Table 5.

3. One exclusion criteria has been added excluding potential subjects with "a history of significant non-adherence or circumstance which would threaten ability to comply with cross-over design and study visit

schedule".

4. Clarified the version of the SF-36 used in this study to be the SF-36v2. All discussion detailing the application of the SF-36 to the study holds true for the SF-36v2.

### Amendment 4 – Addition of blood sample collection for AIM 3 cohort during RHC

In addition to collecting right heart catheter tips, we will collect up to 30 mL (2 tablespoons) of blood at the time of right heart catheterization from all consented subjects enrolled in Aim 3. Platelets and peripheral blood mononuclear cells (PBMCs) will be isolated and analyzed for pathways of metabolomics and for Xist RNA for X chromosome inactivation.

### **Protocol Addendum 1**

Provisions for Study Drug Extension due to COVID-19

For subjects currently enrolled in EDIPHY, we may extend the active treatment period an additional four weeks (Total time of treatment = up to 22 weeks) to complete in person study visits and obtain end points which cannot be obtained virtually/by televisits (i.e., six minute walk distance, cardiac magnetic resonance imaging). This strategy optimizes subject safety (by moving the window out another four weeks, to avoid an in person study visit if conditions so dictate) while minimizing data loss, the chance of "wasted" participation, and our ability to detect efficacy which is best done with a subject on study drug. Based on a prior clinical trial of 381 subjects with systemic lupus erythematosis, which was conducted with a higher dose of DHEA for one year's duration with no serious adverse events (Petri et al., Arthr Rheum 2004), we believe this extension of only four weeks poses no additional risk to subjects.

#### The changes follow:

- 1. Continue study drug until 6MWT and cMRI can be completed (up to an additional 4 weeks); remainder of end points will be assessed virtually on their due date and then coincident with 6MWT and cMRI
- 2. Scheduling
  - a. Active subjects will be contacted proactively to inform them of any relevant updates to study conduct and address any concerns.
  - b. The consent addendum will be sent to their residence and reviewed by phone with a study staff member. If willing, study staff will ask the subject to send the completed form back. Study staff will then sign and send a copy of the consent to the subject.

#### **Visit Procedures**

- 1. Safety Labs and Laboratory Endpoints
  - a. If an off-campus laboratory is available to a subject, safety labs will be drawn and reviewed via remote medical record review.
  - b. Alternatively, if the subject has a previously scheduled clinical visit in the PH Center, safety labs and study labs will be ordered and drawn at this clinic visit.
- 2. 6MWT
  - a. If a subject has a previously scheduled clinical visit in the PH Center, a 6MWT will be performed at this visit.
  - Otherwise, study drug will be continued for up to 4 additional weeks until 6MWT can be obtained
- 3. cMRI
  - a. Study drug will be continued for up to 4 additional weeks until cMRI can be obtained

#### Other Study Drug Details

- 1. Study Drug Dispensing
  - a. Provisions for remote study drug dispensing are being discussed with Lifespan research pharmacy should any subject transition for Period 1 to Period 2.

- b. Research pharmacy will be notified about need for possible additional duration of study drug
- 2. Follow-up in extension period
  - a. Study staff will continue to follow-up and collect adverse events or any other problems the subject may have.
  - b. When a cardiac MRI and 6MWT is able to be scheduled, safety labs will be collected as a "Unscheduled Visit" at this time.
  - c. The Week 19 phone call will occur 1 week after you complete the extension period (if in Treatment Period 1).
  - d. The Week 21 phone call will occur 3 weeks after you complete the extension period (if in Treatment Period 1).
  - e. The Week 42 phone call will occur 2 weeks after you complete the extension period (if in Treatment Period 2).

## **Protocol Addendum 2**

Provisions for COVID-19 Remote Follow-up

In preparation of further COVID-19 precautions, this addendum details provisions to the EDIPHY protocol if remote subject visits become necessary. It seeks to minimize data loss while also ensuring subject safety. Until this point, subject participation will continue per protocol with the addition of ORA/RPO recommended screening procedures.

The changes follow:

#### If remote visits become necessary:

- 1. Continue study drug until 6MWT and cMRI can be completed (up to an additional 4 weeks); remainder of end points will be assessed virtually on their due date and then coincident with 6MWT and cMRI
- 2. Scheduling
  - a. Active subjects will be contacted proactively to inform them of any relevant updates to study conduct and address any concerns.
  - b. If necessary, a remote phone or video visit will be scheduled with the subject.
  - c. The consent addendum will be sent to their residence and reviewed by phone with a study staff member. If willing, study staff will ask the subject to send the completed form back. Study staff will then sign and send a copy of the consent to the subject.

#### **Visit Procedures**

- 1. Safety Labs and Laboratory Endpoints
  - a. If an off-campus laboratory is available to a subject, safety labs will be drawn and reviewed via remote medical record review.
  - b. Alternatively, if the subject has a previously scheduled clinical visit in the PH Center, safety labs and study labs will be ordered and drawn at this clinic visit.
- 2. 6MWT
  - a. If a subject has a previously scheduled clinical visit in the PH Center, a 6MWT will be performed at this visit.
  - Otherwise, study drug will be continued for up to 4 additional weeks until 6MWT can be obtained
- 3. cMRI
  - a. Study drug will be continued for up to 4 additional weeks until cMRI can be obtained
- 4. Quality of Life Surveys
  - a. SF-36v2, emphasis-10 and satisfaction surveys will be administered over the phone and entered directly in REDCap. Alternatively, if the subject feels comfortable, a remote REDCap survey link will be sent to their personal email and completed directly.
- 5. Physician contact

- a. In the absence of an in-person exam, a study physician will remotely perform a review of systems with the subject and assign a WHO functional class at the time of the remote visit.
- 6. Adverse Event, Concomitant Medication and Other Subject Review
  - a. All new or active events, changes in medication and other relevant information will be recorded at the time of the remote visit per standard procedure.
  - b. Study drug adherence will also be reviewed with the subject and recorded.
- 7. Subject Compensation
  - a. A check request form will be completed by study staff and the subject will receive a check commensurate with assigned visit amount within 4-6 weeks.
- 8. Medical Monitor Review
  - a. The independent medical monitor will review all changes necessitated by a shift to remote visits and review the safety information collected per standard procedure.
- 9. Documentation
  - a. Hardcopies of essential study documentation (without PHI) will be brought home with an assigned staff member in preparation for remote visit.
  - b. Documents will be prepared for all active subjects proactively in preparation for any emergent changes.

#### Other

- 1. Study Drug Dispensing
  - a. Provisions for remote study drug dispensing are being discussed with Lifespan research pharmacy should any subject transition for Period 1 to Period 2.
  - b. Research pharmacy will be notified about need for possible additional duration of study drug
- 2. Follow-up in extension period
  - a. Study staff will continue to follow-up and collect adverse events or any other problems the subject may have.
  - b. When a cardiac MRI and 6MWT is able to be scheduled, safety labs will be collected as a "Unscheduled Visit" at this time.
  - c. The Week 42 phone call will now occur 2 weeks after completion of the extension period

## References

- 1. Humbert M, Sitbon O, Chaouat A, Bertocchi M, Habib G, Gressin V, Yaici A, Weitzenblum E, Cordier J-F, Chabot F, Dromer C, Pison C, Reynaud-Gaubert M, Haloun A, Laurent M, Hachulla E, Cottin V, Degano B, Jais X, Montani D, Souza R and Simonneau G. Survival in patients with idiopathic, familial, and anorexigen-associated pulmonary arterial hypertension in the modern management era. *Circulation*. 2010;in press.
- 2. Ventetuolo CE, Ouyang P, Bluemke DA, Tandri H, Barr RG, Bagiella E, Cappola AR, Bristow MR, Johnson C, Kronmal RA, Kizer JR, Lima JA and Kawut SM. Sex Hormones are Associated with Right Ventricular Structure and Function: The MESA-Right Ventricle Study. *Am J Respir Crit Care Med*.201007-1027OC.
- 3. Gabler NB, French B, Strom BL, Liu Z, Palevsky HI, Taichman DB, Kawut SM and Halpern SD. Race and Sex Differences in Response to Endothelin Receptor Antagonists for Pulmonary Arterial Hypertension. *Chest.* 2012;141:20-26.
- 4. Jacobs W, van de Veerdonk MC, Trip P, de Man F, Heymans MW, Marcus JT, Kawut SM, Bogaard HJ, Boonstra A and Vonk Noordegraaf A. The right ventricle explains sex differences in survival in idiopathic pulmonary arterial hypertension. *Chest.* 2014;145:1230-6.
- 5. Ventetuolo CE, Praestgaard A, Palevsky HI, Klinger JR, Halpern SD and Kawut SM. Sex and haemodynamics in pulmonary arterial hypertension. *The European respiratory journal*. 2014;43:523-30.
- 6. Mathai SC, Hassoun PM, Puhan MA, Zhou Y and Wise RA. Gender Differences in Response to Tadalafil in Pulmonary Arterial Hypertension. *Chest*. 2014.
- 7. Meyer P, Filippatos GS, Ahmed MI, Iskandrian AE, Bittner V, Perry GJ, White M, Aban IB, Mujib M, Dell'Italia LJ and Ahmed A. Effects of right ventricular ejection fraction on outcomes in chronic systolic heart Version date 8/12/2021

failure. Circulation. 2010;121:252-8.

- 8. Mohammed SF, Hussain I, Abou Ezzeddine OF, Takahama H, Kwon SH, Forfia P, Roger VL and Redfield MM. Right ventricular function in heart failure with preserved ejection fraction: a community-based study. *Circulation*. 2014;130:2310-20.
- 9. Morrison DA, Adcock K, Collins CM, Goldman S, Caldwell JH and Schwarz MI. Right ventricular dysfunction and the exercise limitation of chronic obstructive pulmonary disease. *Journal of the American College of Cardiology*. 1987;9:1219-29.
- 10. D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Kernis JT and et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. *Ann Intern Med*. 1991;115:343-9.
- 11. Lahm T, Tuder RM and Petrache I. Progress in solving the sex hormone paradox in pulmonary hypertension. *American journal of physiology Lung cellular and molecular physiology*. 2014;307:L7-26.
- 12. Benza RL, Miller DP, Gomberg-Maitland M, Frantz RP, Foreman AJ, Coffey CS, Frost A, Barst RJ, Badesch DB, Elliott CG, Liou TG and McGoon MD. Predicting Survival in Pulmonary Arterial Hypertension. Insights From the Registry to Evaluate Early and Long-Term Pulmonary Arterial Hypertension Disease Management (REVEAL). *Circulation*.CIRCULATIONAHA.109.898122.
- 13. Ventetuolo CE, Baird GL, Barr RG, Bluemke DA, Fritz JS, Hill NS, Klinger JR, Lima JA, Ouyang P, Palevsky HI, Palmisciano AJ, Krishnan I, Pinder D, Preston IR, Roberts KE and Kawut SM. Higher Estradiol and Lower Dehydroepiandrosterone-Sulfate Levels Are Associated with Pulmonary Arterial Hypertension in Men. *American journal of respiratory and critical care medicine*. 2016;193:1168-75.
- 14. Kawut SM, Archer-Chicko CL, DeMichele A, Fritz JS, Klinger JR, Ky B, Palevsky HI, Palmisciano AJ, Patel M, Pinder D, Propert KJ, Smith KA, Stanczyk F, Tracy R, Vaidya A, Whittenhall ME and Ventetuolo CE. Anastrozole in Pulmonary Arterial Hypertension. A Randomized, Double-Blind, Placebo-controlled Trial. *American journal of respiratory and critical care medicine*. 2017;195:360-368.
- 15. Bonnet S, Dumas-de-La-Roque E, Begueret H, Marthan R, Fayon M, Dos Santos P, Savineau J and Baulieu E. Dehydroepiandrosterone (DHEA) prevents and reverses chronic hypoxic pulmonary hypertension. *Proc Natl Acad Sci USA*. 2003;100:9488 9493.
- 16. Hampl V, Bibova J, Povysilova V and Herget J. Dehydroepiandrosterone sulphate reduces chronic hypoxic pulmonary hypertension in rats. *The European respiratory journal*. 2003;21:862 865.
- 17. Dumas de La Roque E, Bellance N, Rossignol R, Begueret H, Billaud M, dos Santos P, Ducret T, Marthan R, Dahan D, Ramos-Barbon D, Amor-Carro O, Savineau JP and Fayon M. Dehydroepiandrosterone reverses chronic hypoxia/reoxygenation-induced right ventricular dysfunction in rats. *The European respiratory journal*. 2012;40:1420-9.
- 18. Alzoubi A, Toba M, Abe K, O'Neill KD, Rocic P, Fagan KA, McMurtry IF and Oka M. Dehydroepiandrosterone restores right ventricular structure and function in rats with severe pulmonary arterial hypertension. *American journal of physiology Heart and circulatory physiology*. 2013;304:H1708-18.
- 19. Paulin R, Meloche J, Jacob MH, Bisserier M, Courboulin A and Bonnet S. Dehydroepiandrosterone inhibits the Src/STAT3 constitutive activation in pulmonary arterial hypertension. *American journal of physiology Heart and circulatory physiology*. 2011;301:H1798-809.
- 20. Nakamura S, Yoshimura M, Nakayama M, Ito T, Mizuno Y, Harada E, Sakamoto T, Saito Y, Nakao K, Yasue H and Ogawa H. Possible association of heart failure status with synthetic balance between aldosterone and dehydroepiandrosterone in human heart. *Circulation*. 2004;110:1787-93.
- 21. Mannic T, Mouffok M, Python M, Yoshida T, Maturana AD, Vuilleumier N and Rossier MF. DHEA prevents mineralo- and glucocorticoid receptor-induced chronotropic and hypertrophic actions in isolated rat cardiomyocytes. *Endocrinology*. 2013;154:1271-81.
- 22. Liu D and Dillon JS. Dehydroepiandrosterone Activates Endothelial Cell Nitric-oxide Synthase by a Specific Plasma Membrane Receptor Coupled to Gαi2,3. *Journal of Biological Chemistry*. 2002;277:21379-21388.
- 23. Chen H, Lin AS, Li Y, Reiter CEN, Ver MR and Quon MJ. Dehydroepiandrosterone Stimulates Phosphorylation of FoxO1 in Vascular Endothelial Cells via Phosphatidylinositol 3-Kinase- and Protein Kinase A-dependent Signaling Pathways to Regulate ET-1 Synthesis and Secretion. *Journal of Biological Chemistry*. 2008;283:29228-29238.
- 24. Forte P, Kneale BJ, Milne E, Chowienczyk PJ, Johnston A, Benjamin N and Ritter JM. Evidence for a difference in nitric oxide biosynthesis between healthy women and men. *Hypertension*. 1998;32:730-4.
- 25. Davidge ST, Stranko CP and Roberts JM. Urine but not plasma nitric oxide metabolites are decreased

in women with preeclampsia. American journal of obstetrics and gynecology. 1996;174:1008-13.

- 26. Stauffer BL, Westby CM, Greiner JJ, Van Guilder GP and Desouza CA. Sex differences in endothelin-1-mediated vasoconstrictor tone in middle-aged and older adults. *American journal of physiology Regulatory, integrative and comparative physiology.* 2010;298:R261-5.
- 27. Polderman KH, Stehouwer CD, van Kamp GJ, Dekker GA, Verheugt FW and Gooren LJ. Influence of sex hormones on plasma endothelin levels. *Annals of internal medicine*. 1993;118:429-32.
- 28. Miyauchi T, Yanagisawa M, Iida K, Ajisaka R, Suzuki N, Fujino M, Goto K, Masaki T and Sugishita Y. Age- and sex-related variation of plasma endothelin-1 concentration in normal and hypertensive subjects. *American heart journal*. 1992;123:1092-3.
- 29. Sasaki H, Nagayama T, Blanton RM, Seo K, Zhang M, Zhu G, Lee DI, Bedja D, Hsu S, Tsukamoto O, Takashima S, Kitakaze M, Mendelsohn ME, Karas RH, Kass DA and Takimoto E. PDE5 inhibitor efficacy is estrogen dependent in female heart disease. *The Journal of clinical investigation*. 2014;124:2464-71.
- 30. Badesch DB, Raskob GE, Elliott CG, Krichman AM, Farber HW, Frost AE, Barst RJ, Benza RL, Liou TG, Turner M, Giles S, Feldkircher K, Miller DP and McGoon MD. Pulmonary Arterial Hypertension: Baseline characteristics from the REVEAL registry. *Chest*. 2010;137:376-387.
- 31. Benza RL, Miller DP, Gomberg-Maitland M, Frantz RP, Foreman AJ, Coffey CS, Frost A, Barst RJ, Badesch DB, Elliott CG, Liou TG and McGoon MD. Predicting Survival in Pulmonary Arterial Hypertension: Insights From the Registry to Evaluate Early and Long-Term Pulmonary Arterial Hypertension Disease Management (REVEAL). *Circulation*. 122:164-172.
- 32. Kawut SM, Lima JAC, Barr RG, Chahal H, Jain A, Tandri H, Praestgaard A, Bagiella E, Kizer JR, Johnson WC, Kronmal RA and Bluemke DA. Sex and Race Differences in Right Ventricular Structure and Function: The Multi-Ethnic Study of Atherosclerosis-Right Ventricle Study. *Circulation*. 123:2542-2551.
- 33. Melenovsky V, Hwang SJ, Lin G, Redfield MM and Borlaug BA. Right heart dysfunction in heart failure with preserved ejection fraction. *European heart journal*. 2014;35:3452-62.
- 34. Kawut SM, Al-Naamani N, Agerstrand C, Berman Rosenzweig E, Rowan C, Barst RJ, Bergmann S and Horn EM. Determinants of Right Ventricular Ejection Fraction in Pulmonary Arterial Hypertension. *Chest*. 2009:135:752-759.
- 35. Peacock AJ, Crawley S, McLure L, Blyth K, Vizza CD, Poscia R, Francone M, Iacucci I, Olschewski H, Kovacs G, Vonk Noordegraaf A, Marcus JT, van de Veerdonk MC and Oosterveer FP. Changes in right ventricular function measured by cardiac magnetic resonance imaging in patients receiving pulmonary arterial hypertension-targeted therapy: the EURO-MR study. *Circulation Cardiovascular imaging*. 2014;7:107-14.
- 36. Dumas de la Roque E, Quignard JF, Ducret T, Dahan D, Courtois A, Begueret H, Marthan R and Savineau JP. Beneficial effect of dehydroepiandrosterone on pulmonary hypertension in a rodent model of pulmonary hypertension in infants. *Pediatric research*. 2013;74:163-9.
- 37. Oka M, Karoor V, Homma N, Nagaoka T, Sakao E, Golembeski SM, Limbird J, Imamura M, Gebb SA, Fagan KA and McMurtry IF. Dehydroepiandrosterone upregulates soluble guanylate cyclase and inhibits hypoxic pulmonary hypertension. *Cardiovascular research*. 2007;74:377-87.
- 38. Homma N, Nagaoka T, Karoor V, Imamura M, Taraseviciene-Stewart L, Walker LA, Fagan KA, McMurtry IF and Oka M. Involvement of RhoA/Rho kinase signaling in protection against monocrotaline-induced pulmonary hypertension in pneumonectomized rats by dehydroepiandrosterone. *American journal of physiology Lung cellular and molecular physiology*. 2008;295:L71-78.
- 39. White K, Johansen AK, Nilsen M, Ciuclan L, Wallace E, Paton L, Campbell A, Morecroft I, Loughlin L, McClure JD, Thomas M, Mair KM and MacLean MR. Activity of the estrogen-metabolizing enzyme cytochrome P450 1B1 influences the development of pulmonary arterial hypertension. *Circulation*. 2012;126:1087-98.
- 40. Akishita M, Hashimoto M, Ohike Y, Ogawa S, Iijima K, Eto M and Ouchi Y. Association of plasma dehydroepiandrosterone-sulfate levels with endothelial function in postmenopausal women with coronary risk factors. *Hypertension research : official journal of the Japanese Society of Hypertension*. 2008;31:69-74.
- 41. Kawano H, Yasue H, Kitagawa A, Hirai N, Yoshida T, Soejima H, Miyamoto S, Nakano M and Ogawa H. Dehydroepiandrosterone supplementation improves endothelial function and insulin sensitivity in men. *The Journal of clinical endocrinology and metabolism*. 2003;88:3190-5.
- 42. Barrett-Connor E, Khaw KT and Yen SS. A prospective study of dehydroepiandrosterone sulfate, mortality, and cardiovascular disease. *The New England journal of medicine*. 1986;315:1519-24.
- 43. Shufelt C, Bretsky P, Almeida CM, Johnson BD, Shaw LJ, Azziz R, Braunstein GD, Pepine CJ, Bittner V, Vido DA, Stanczyk FZ and Bairey Merz CN. DHEA-S levels and cardiovascular disease mortality in postmenopausal women: results from the National Institutes of Health--National Heart, Lung, and Blood

- Institute (NHLBI)-sponsored Women's Ischemia Syndrome Evaluation (WISE). *The Journal of clinical endocrinology and metabolism*. 2010;95:4985-92.
- 44. Herrington DM. Dehydroepiandrosterone and coronary atherosclerosis. *Annals of the New York Academy of Sciences*. 1995;774:271-80.
- 45. Feldman HA, Johannes CB, Araujo AB, Mohr BA, Longcope C and McKinlay JB. Low dehydroepiandrosterone and ischemic heart disease in middle-aged men: prospective results from the Massachusetts Male Aging Study. *American journal of epidemiology*. 2001;153:79-89.
- 46. Moriyama Y, Yasue H, Yoshimura M, Mizuno Y, Nishiyama K, Tsunoda R, Kawano H, Kugiyama K, Ogawa H, Saito Y and Nakao K. The plasma levels of dehydroepiandrosterone sulfate are decreased in patients with chronic heart failure in proportion to the severity. *The Journal of clinical endocrinology and metabolism.* 2000;85:1834-40.
- 47. Aragno M, Mastrocola R, Alloatti G, Vercellinatto I, Bardini P, Geuna S, Catalano MG, Danni O and Boccuzzi G. Oxidative stress triggers cardiac fibrosis in the heart of diabetic rats. *Endocrinology*. 2008;149:380-8.
- 48. Aragno M, Meineri G, Vercellinatto I, Bardini P, Raimondo S, Peiretti PG, Vercelli A, Alloatti G, Tomasinelli CE, Danni O and Boccuzzi G. Cardiac impairment in rabbits fed a high-fat diet is counteracted by dehydroepiandrosterone supplementation. *Life sciences*. 2009;85:77-84.
- 49. Rain S, Andersen S, Najafi A, Gammelgaard Schultz J, da Silva Goncalves Bos D, Handoko ML, Bogaard HJ, Vonk-Noordegraaf A, Andersen A, van der Velden J, Ottenheijm CA and de Man FS. Right Ventricular Myocardial Stiffness in Experimental Pulmonary Arterial Hypertension: Relative Contribution of Fibrosis and Myofibril Stiffness. *Circulation Heart failure*. 2016;9.
- Nagendran J, Sutendra G, Paterson I, Champion HC, Webster L, Chiu B, Haromy A, Rebeyka IM, Ross DB and Michelakis ED. Endothelin Axis Is Upregulated in Human and Rat Right Ventricular Hypertrophy. *Circulation Research*. 2013;112:347-354.
- 51. Sandstede J, Lipke C, Beer M, Hofmann S, Pabst T, Kenn W, Neubauer S and Hahn D. Age- and gender-specific differences in left and right ventricular cardiac function and mass determined by cine magnetic resonance imaging. *Eur Radiol*. 2000;10:438-42.
- 52. Grothues F, Moon JC, Bellenger NG, Smith GS, Klein HU and Pennell DJ. Interstudy reproducibility of right ventricular volumes, function, and mass with cardiovascular magnetic resonance. *Am Heart J*. 2004:147:218-23.
- 53. Beygui F, Furber A, Delépine S, Helft G, Metzger J-P, Geslin P and Jeune J. Routine breath-hold gradient echo MRI-derived right ventricular mass, volumes and function: accuracy, reproducibility and coherence study. *The International Journal of Cardiovascular Imaging (formerly Cardiac Imaging)*. 2004;20:509-516.
- 54. Kawut SM, Barr RG, Lima JAC, Praestgaard A, Johnson WC, Chahal H, Ogunyankin KO, Bristow MR, Kizer JR, Tandri H and Bluemke DA. Right Ventricular Structure Is Associated With the Risk of Heart Failure and Cardiovascular Death: The Multi-Ethnic Study of Atherosclerosis (MESA)-Right Ventricle Study. *Circulation*. 2012;126:1681-1688.
- 55. Hardegree EL, Sachdev A, Villarraga HR, Frantz RP, McGoon MD, Kushwaha SS, Hsiao JF, McCully RB, Oh JK, Pellikka PA and Kane GC. Role of serial quantitative assessment of right ventricular function by strain in pulmonary arterial hypertension. *Am J Cardiol*. 2013;111:143-8.
- 56. Sachdev A, Villarraga HR, Frantz RP, McGoon MD, Hsiao JF, Maalouf JF, Ammash NM, McCully RB, Miller FA, Pellikka PA, Oh JK and Kane GC. Right ventricular strain for prediction of survival in patients with pulmonary arterial hypertension. *Chest.* 2011;139:1299-309.
- 57. Ohyama Y, Ambale-Venkatesh B, Chamera E, Shehata ML, Corona-Villalobos CP, Zimmerman SL, Hassoun PM, Bluemke DA and Lima JA. Comparison of strain measurement from multimodality tissue tracking with strain-encoding MRI and harmonic phase MRI in pulmonary hypertension. *International journal of cardiology*. 2015;182:342-8.
- 58. van Wolferen SA, van de Veerdonk MC, Mauritz G-J, Jacobs W, Marcus JT, Marques KMJ, Bronzwaer JGF, Heymans MW, Boonstra A, Postmus PE, Westerhof N and Vonk Noordegraaf A. Clinically Significant Change in Stroke Volume in Pulmonary Hypertension. *Chest*. 2011;139:1003-1009.
- 59. van Wolferen SA, Marcus JT, Boonstra A, Marques KM, Bronzwaer JG, Spreeuwenberg MD, Postmus PE and Vonk-Noordegraaf A. Prognostic value of right ventricular mass, volume, and function in idiopathic pulmonary arterial hypertension. *European heart journal*. 2007;28:1250-7.
- 60. van de Veerdonk MC, Kind T, Marcus JT, Mauritz GJ, Heymans MW, Bogaard HJ, Boonstra A,

- Marques KM, Westerhof N and Vonk-Noordegraaf A. Progressive right ventricular dysfunction in patients with pulmonary arterial hypertension responding to therapy. *Journal of the American College of Cardiology*. 2011;58:2511-9.
- 61. Calvier L, Legchenko E, Grimm L, Sallmon H, Hatch A, Plouffe BD, Schroeder C, Bauersachs J, Murthy SK and Hansmann G. Galectin-3 and aldosterone as potential tandem biomarkers in pulmonary arterial hypertension. *Heart (British Cardiac Society)*. 2016;102:390-6.
- 62. Fenster BE, Lasalvia L, Schroeder JD, Smyser J, Silveira LJ, Buckner JK and Brown KK. Galectin-3 levels are associated with right ventricular functional and morphologic changes in pulmonary arterial hypertension. *Heart and vessels*. 2016;31:939-46.
- 63. Suzuki S, Nakazato K, Sugimoto K, Yoshihisa A, Yamaki T, Kunii H, Suzuki H, Saitoh S and Takeishi Y. Plasma Levels of Receptor for Advanced Glycation End-Products and High-Mobility Group Box 1 in Patients With Pulmonary Hypertension. *International heart journal*. 2016;57:234-40.
- 64. Meloche J, Courchesne A, Barrier M, Carter S, Bisserier M, Paulin R, Lauzon-Joset JF, Breuils-Bonnet S, Tremblay E, Biardel S, Racine C, Courture C, Bonnet P, Majka SM, Deshaies Y, Picard F, Provencher S and Bonnet S. Critical role for the advanced glycation end-products receptor in pulmonary arterial hypertension etiology. *Journal of the American Heart Association*. 2013;2:e005157.
- 65. Jiang X, Guo CX, Zeng XJ, Li HH, Chen BX and Du FH. A soluble receptor for advanced glycation end-products inhibits myocardial apoptosis induced by ischemia/reperfusion via the JAK2/STAT3 pathway. *Apoptosis : an international journal on programmed cell death*. 2015;20:1033-47.
- 66. Meuwese MC, Stroes ES, Hazen SL, van Miert JN, Kuivenhoven JA, Schaub RG, Wareham NJ, Luben R, Kastelein JJ, Khaw KT and Boekholdt SM. Serum myeloperoxidase levels are associated with the future risk of coronary artery disease in apparently healthy individuals: the EPIC-Norfolk Prospective Population Study. *Journal of the American College of Cardiology*. 2007;50:159-65.
- 67. Brennan M-L, Penn MS, Van Lente F, Nambi V, Shishehbor MH, Aviles RJ, Goormastic M, Pepoy ML, McErlean ES, Topol EJ, Nissen SE and Hazen SL. Prognostic Value of Myeloperoxidase in Patients with Chest Pain. *New England Journal of Medicine*. 2003;349:1595-1604.
- 68. Schindhelm RK, van der Zwan LP, Teerlink T and Scheffer PG. Myeloperoxidase: a useful biomarker for cardiovascular disease risk stratification? *Clinical chemistry*. 2009;55:1462-70.
- 69. Niccoli G, Celestini A, Calvieri C, Cosentino N, Falcioni E, Carnevale R, Nocella C, Fracassi F, Roberto M, Antonazzo RP, Pignatelli P, Crea F and Violi F. Patients with microvascular obstruction after primary percutaneous coronary intervention show a gp91phox (NOX2) mediated persistent oxidative stress after reperfusion. *European heart journal Acute cardiovascular care*. 2013;2:379-88.
- 70. Loffredo L, Martino F, Carnevale R, Pignatelli P, Catasca E, Perri L, Calabrese CM, Palumbo MM, Baratta F, Del Ben M, Angelico F and Violi F. Obesity and hypercholesterolemia are associated with NOX2 generated oxidative stress and arterial dysfunction. *The Journal of pediatrics*. 2012;161:1004-9.
- 71. Pignatelli P, Carnevale R, Cangemi R, Loffredo L, Sanguigni V, Stefanutti C, Basili S and Violi F. Atorvastatin inhibits gp91phox circulating levels in patients with hypercholesterolemia. *Arteriosclerosis, thrombosis, and vascular biology.* 2010;30:360-7.
- 72. Weiss EP, Villareal DT, Ehsani AA, Fontana L and Holloszy JO. Dehydroepiandrosterone replacement therapy in older adults improves indices of arterial stiffness. *Aging cell*. 2012;11:876-84.
- 73. Soon E, Holmes AM, Treacy CM, Doughty NJ, Southgate L, Machado RD, Trembath RC, Jennings S, Barker L, Nicklin P, Walker C, Budd DC, Pepke-Zaba J and Morrell NW. Elevated levels of inflammatory cytokines predict survival in idiopathic and familial pulmonary arterial hypertension. *Circulation*. 2010;122:920-7.
- 74. Matura LA, Ventetuolo CE, Palevsky HI, Lederer DJ, Horn EM, Mathai SC, Pinder D, Archer-Chicko C, Bagiella E, Roberts KE, Tracy RP, Hassoun PM, Girgis RE and Kawut SM. Interleukin-6 and tumor necrosis factor-alpha are associated with quality of life-related symptoms in pulmonary arterial hypertension. *Annals of the American Thoracic Society*. 2015;12:370-5.
- 75. Alkatib AA, Cosma M, Elamin MB, Erickson D, Swiglo BA, Erwin PJ and Montori VM. A systematic review and meta-analysis of randomized placebo-controlled trials of DHEA treatment effects on quality of life in women with adrenal insufficiency. *The Journal of clinical endocrinology and metabolism*. 2009;94:3676-81.
- 76. Crosbie D, Black C, McIntyre L, Royle PL and Thomas S. Dehydroepiandrosterone for systemic lupus erythematosus. *The Cochrane database of systematic reviews*. 2007:Cd005114.
- 77. Petri MA, Mease PJ, Merrill JT, Lahita RG, Iannini MJ, Yocum DE, Ginzler EM, Katz RS, Gluck OS, Genovese MC, Van Vollenhoven R, Kalunian KC, Manzi S, Greenwald MW, Buyon JP, Olsen NJ, Schiff MH,

- Kavanaugh AF, Caldwell JR, Ramsey-Goldman R, St Clair EW, Goldman AL, Egan RM, Polisson RP, Moder KG, Rothfield NF, Spencer RT, Hobbs K, Fessler BJ, Calabrese LH, Moreland LW, Cohen SB, Quarles BJ, Strand V, Gurwith M and Schwartz KE. Effects of prasterone on disease activity and symptoms in women with active systemic lupus erythematosus. *Arthritis and rheumatism*. 2004;50:2858-68.
- 78. Dumas de La Roque E, Savineau JP, Metivier AC, Billes MA, Kraemer JP, Doutreleau S, Jougon J, Marthan R, Moore N, Fayon M, Baulieu EE and Dromer C. Dehydroepiandrosterone (DHEA) improves pulmonary hypertension in chronic obstructive pulmonary disease (COPD): a pilot study. *Annales d'endocrinologie*. 2012;73:20-5.
- 79. Wang L, Hao Q, Wang YD, Wang WJ and Li DJ. Protective effects of dehydroepiandrosterone on atherosclerosis in ovariectomized rabbits via alleviating inflammatory injury in endothelial cells. *Atherosclerosis*. 2011;214:47-57.
- 80. Lee MJ, Kim EH, Lee SA, Kang YM, Jung CH, Yoon HK, Seol SM, Lee YL, Lee WJ and Park JY. Dehydroepiandrosterone prevents linoleic acid-induced endothelial cell senescence by increasing autophagy. *Metabolism: clinical and experimental.* 2015;64:1134-45.
- 81. Huerta-Garcia E, Ventura-Gallegos JL, Victoriano ME, Montiel-Davalos A, Tinoco-Jaramillo G and Lopez-Marure R. Dehydroepiandrosterone inhibits the activation and dysfunction of endothelial cells induced by high glucose concentration. *Steroids*. 2012;77:233-40.
- 82. Barkhausen T, Westphal BM, Putz C, Krettek C and van Griensven M. Dehydroepiandrosterone administration modulates endothelial and neutrophil adhesion molecule expression in vitro. *Critical care (London, England)*. 2006;10:R109.
- 83. Altman R, Motton DD, Kota RS and Rutledge JC. Inhibition of vascular inflammation by dehydroepiandrosterone sulfate in human aortic endothelial cells: roles of PPARalpha and NF-kappaB. *Vascular pharmacology*. 2008;48:76-84.
- 84. Milewich L, Hendricks TS and Johnson AR. Metabolism of dehydroisoandrosterone and androstenedione in human pulmonary endothelial cells in culture. *The Journal of clinical endocrinology and metabolism*. 1983;56:930-5.
- 85. Shapiro S, Traiger GL, Turner M, McGoon MD, Wason P and Barst RJ. Sex Differences in the Diagnosis, Treatment, and Outcome of Patients With Pulmonary Arterial Hypertension Enrolled in the Registry to Evaluate Early and Long-term Pulmonary Arterial Hypertension Disease ManagementSex Differences in Pulmonary Arterial Hypertension. *CHEST Journal*. 2012;141:363-373.
- 86. Roberts KE, Fallon MB, Krowka MJ, Brown RS, Trotter JF, Peter I, Tighiouart H, Knowles JA, Rabinowitz D, Benza RL, Badesch DB, Taichman DB, Horn EM, Zacks S, Kaplowitz N and Kawut SM. Genetic risk factors for portopulmonary hypertension in patients with advanced liver disease. *American journal of respiratory and critical care medicine*. 2009;179:835-42.
- 87. Austin ED, Cogan JD, West JD, Hedges LK, Hamid R, Dawson EP, Wheeler LA, Parl FF, Loyd JE and Phillips JA. Alterations in oestrogen metabolism: implications for higher penetrance of familial pulmonary arterial hypertension in females. *European Respiratory Journal*. 2009;34:1093-1099.
- 88. Russell KS, Haynes MP, Sinha D, Clerisme E and Bender JR. Human vascular endothelial cells contain membrane binding sites for estradiol, which mediate rapid intracellular signaling. *Proceedings of the National Academy of Sciences of the United States of America*. 2000;97:5930-5.
- 89. Billon-Gales A, Fontaine C, Filipe C, Douin-Echinard V, Fouque MJ, Flouriot G, Gourdy P, Lenfant F, Laurell H, Krust A, Chambon P and Arnal JF. The transactivating function 1 of estrogen receptor alpha is dispensable for the vasculoprotective actions of 17beta-estradiol. *Proceedings of the National Academy of Sciences of the United States of America*. 2009;106:2053-8.
- 90. White K, Dempsie Y, Nilsen M, Wright AF, Loughlin L and MacLean MR. The serotonin transporter, gender, and 17β oestradiol in the development of pulmonary arterial hypertension. *Cardiovascular research*. 2011;90:373-382.
- 91. Dempsie Y, Nilsen M, White K, Mair KM, Loughlin L, Ambartsumian N, Rabinovitch M and MacLean MR. Development of pulmonary arterial hypertension in mice over-expressing S100A4/Mts1 is specific to females. *Respiratory research*. 2011;12:159-159.
- 92. Dempsie Y, MacRitchie NA, White K, Morecroft I, Wright AF, Nilsen M, Loughlin L, Mair KM and MacLean MR. Dexfenfluramine and the oestrogen-metabolizing enzyme CYP1B1 in the development of pulmonary arterial hypertension. *Cardiovascular research*. 2013;99:24-34.
- 93. Lahm T, Patel KM, Crisostomo PR, Markel TA, Wang M, Herring C and Meldrum DR. Endogenous estrogen attenuates pulmonary artery vasoreactivity and acute hypoxic pulmonary vasoconstriction: the effects

- of sex and menstrual cycle. *American Journal of Physiology Endocrinology and Metabolism*. 2007;293:E865-E871.
- 94. Kirson NY, Birnbaum HG, Ivanova JI, Waldman T, Joish V and Williamson T. Excess costs associated with patients with chronic thromboembolic pulmonary hypertension in a US privately insured population. *Appl Health Econ Health Policy*. 2011;9:377-87.
- 95. Copher R, Cerulli A, Watkins A and Laura Monsalvo M. Treatment patterns and healthcare system burden of managed care patients with suspected pulmonary arterial hypertension in the United States. *J Med Econ.* 2012;15:947-55.
- 96. Galie N, Barbera JA, Frost AE, Ghofrani HA, Hoeper MM, McLaughlin VV, Peacock AJ, Simonneau G, Vachiery JL, Grunig E, Oudiz RJ, Vonk-Noordegraaf A, White RJ, Blair C, Gillies H, Miller KL, Harris JH, Langley J and Rubin LJ. Initial Use of Ambrisentan plus Tadalafil in Pulmonary Arterial Hypertension. *The New England journal of medicine*. 2015;373:834-44.
- 97. Erzurum S, Rounds SI, Stevens T, Aldred M, Aliotta J, Archer SL, Asosingh K, Balaban R, Bauer N, Bhattacharya J, Bogaard HJ, Choudhary G, Dorn II GW, Dweik R, Fagan K, Fallon M, Finkel T, Geraci M, Gladwin MT, Hassoun PM, Humbert M, Kaminski N, Kawut SM, Loscalzo J, McDonald D, McMurtry IF, Newman J, Nicolls M, Rabinovitch M, Shizuru J, Oka M, Polgar P, Rodman D, Schumacker P, Stenmark K, Tuder R, Voelkel NF, Sullivan E, Weinshilboum R, Yoder MC, Zhao Y, Gail D and Moore TM. Strategic Plan for Lung Vascular Research: An NHLBI-ORDR Workshop Report. *Am J Respir Crit Care Med*.201006-0869WS.
- 98. Newman JH, Rich S, Abman SH, Alexander JH, Barnard J, Beck GJ, Benza RL, Bull TM, Chan SY, Chun HJ, Doogan D, Dupuis J, Erzurum SC, Frantz RP, Geraci M, Gillies H, Gladwin M, Gray MP, Hemnes AR, Herbst RS, Hernandez AF, Hill NS, Horn EM, Hunter K, Jing ZC, Johns R, Kaul S, Kawut SM, Lahm T, Leopold JA, Lewis GD, Mathai SC, McLaughlin VV, Michelakis ED, Nathan SD, Nichols W, Page G, Rabinovitch M, Rich J, Rischard F, Rounds S, Shah SJ, Tapson VF, Lowy N, Stockbridge N, Weinmann G and Xiao L. Enhancing Insights into Pulmonary Vascular Disease (PVD) Through a Precision Medicine Approach. A Joint NHLBI-CMREF Workshop Report. *American journal of respiratory and critical care medicine*. 2017.
- 99. Ventetuolo CE, Baird GL, Barr RG, Bluemke DA, Fritz JS, Hill NS, Klinger JR, Lima JA, Ouyang P, Palevsky HI, Palmisciano AJ, Krishnan I, Pinder D, Preston IR, Roberts KE and Kawut SM. Higher Estradiol and Lower Dehydroepiandrosterone-Sulfate Levels Are Associated With Pulmonary Arterial Hypertension in Men. *American journal of respiratory and critical care medicine*. 2015.
- 100. Pollett JB, Benza RL, Murali S, Shields KJ and Passineau MJ. Harvest of pulmonary artery endothelial cells from patients undergoing right heart catheterization. *The Journal of heart and lung transplantation : the official publication of the International Society for Heart Transplantation*. 2013;32:746-9.
- 101. Zhao X-J, Wang L, Shiva S, Tejero J, Myerburg MM, Wang J, Frizzell S and Gladwin MT. Mechanisms for cellular NO oxidation and nitrite formation in lung epithelial cells. *Free Radical Biology and Medicine*. 2013;61:428-437.
- 102. Zuckerbraun BS, Shiva S, Ifedigbo E, Mathier MA, Mollen KP, Rao J, Bauer PM, Choi JJ, Curtis E, Choi AM and Gladwin MT. Nitrite potently inhibits hypoxic and inflammatory pulmonary arterial hypertension and smooth muscle proliferation via xanthine oxidoreductase-dependent nitric oxide generation. *Circulation*. 2010;121:98-109.
- 103. Aliotta JM, Pereira M, Amaral A, Sorokina A, Igbinoba Z, Hasslinger A, El-Bizri R, Rounds SI, Quesenberry PJ and Klinger JR. Induction of pulmonary hypertensive changes by extracellular vesicles from monocrotaline-treated mice. *Cardiovascular research*. 2013;100:354-362.
- 104. Aliotta JM, Keaney PJ, Warburton RR, DelTatto M, Dooner MS, Passero MA, Quesenberry PJ and Klinger JR. Marrow Cell Infusion Attenuates Vascular Remodeling in a Murine Model of Monocrotaline-Induced Pulmonary Hypertension. *Stem Cells and Development*. 2009;18:773-781.
- 105. Aliotta JM, Passero M, Meharg J, Klinger J, Dooner MS, Pimentel J and Quesenberry PJ. Stem cells and pulmonary metamorphosis: New concepts in repair and regeneration. *Journal of Cellular Physiology*. 2005;204:725-741.
- 106. Aliotta JM, Pereira M, Wen S, Dooner MS, Del Tatto M, Papa E, Goldberg LR, Baird GL, Ventetuolo CE, Quesenberry PJ and Klinger JR. Exosomes induce and reverse monocrotaline-induced pulmonary hypertension in mice. *Cardiovascular research*. 2016;110:319-30.
- 107. Arlt W, Callies F, van Vlijmen JC, Koehler I, Reincke M, Bidlingmaier M, Huebler D, Oettel M, Ernst M, Schulte HM and Allolio B. Dehydroepiandrosterone replacement in women with adrenal insufficiency. *The New England journal of medicine*. 1999:341:1013-20.
- 108. Arlt W, Justl HG, Callies F, Reincke M, Hubler D, Oettel M, Ernst M, Schulte HM and Allolio B. Oral

- dehydroepiandrosterone for adrenal androgen replacement: pharmacokinetics and peripheral conversion to androgens and estrogens in young healthy females after dexamethasone suppression. *The Journal of clinical endocrinology and metabolism*. 1998;83:1928-34.
- 109. Wilkins MR, Paul GA, Strange JW, Tunariu N, Gin-Sing W, Banya WA, Westwood MA, Stefanidis A, Ng LL, Pennell DJ, Mohiaddin RH, Nihoyannopoulos P and Gibbs JS. Sildenafil versus Endothelin Receptor Antagonist for Pulmonary Hypertension (SERAPH) study. *American journal of respiratory and critical care medicine*. 2005;171:1292-7.
- 110. Gan CT, Holverda S, Marcus JT, Paulus WJ, Marques KM, Bronzwaer JG, Twisk JW, Boonstra A, Postmus PE and Vonk-Noordegraaf A. Right ventricular diastolic dysfunction and the acute effects of sildenafil in pulmonary hypertension patients. *Chest.* 2007;132:11-7.
- 111. Natori S, Lai S, Finn JP, Gomes AS, Hundley WG, Jerosch-Herold M, Pearson G, Sinha S, Arai A, Lima JAC and Bluemke DA. Cardiovascular Function in Multi-Ethnic Study of Atherosclerosis: Normal Values by Age, Sex, and Ethnicity. *Am J Roentgenol*. 2006;186:S357-365.
- 112. Leuchte HH, El Nounou M, Tuerpe JC, Hartmann B, Baumgartner RA, Vogeser M, Muehling O and Behr J. N-terminal pro-brain natriuretic peptide and renal insufficiency as predictors of mortality in pulmonary hypertension. *Chest*. 2007;131:402-9.
- 113. Souza R, Bogossian HB, Humbert M, Jardim C, Rabelo R, Amato MB and Carvalho CR. N-terminal-pro-brain natriuretic peptide as a haemodynamic marker in idiopathic pulmonary arterial hypertension. *The European respiratory journal*. 2005;25:509-13.
- 114. Chen H, De Marco T, Kobashigawa EA, Katz PP, Chang VW and Blanc PD. Comparison of cardiac and pulmonary-specific quality-of-life measures in pulmonary arterial hypertension. *The European respiratory journal*. 2011;38:608-16.
- 115. McHorney CA, Ware JE, Jr., Lu JF and Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. *Medical care*. 1994;32:40-66.
- 116. Pepke-Zaba J, Beardsworth A, Chan M and Angalakuditi M. Tadalafil therapy and health-related quality of life in pulmonary arterial hypertension. *Current medical research and opinion*. 2009;25:2479-85.
- 117. Pepke-Zaba J, Gilbert C, Collings L and Brown MC. Sildenafil improves health-related quality of life in patients with pulmonary arterial hypertension. *Chest*. 2008;133:183-9.
- 118. Mathai SC, Suber T, Khair RM, Kolb TM, Damico RL and Hassoun PM. Health-Related Quality of Life and Survival in Pulmonary Arterial Hypertension. *Annals of the American Thoracic Society*. 2015.
- 119. Fernandes CJ, Martins BC, Jardim CV, Ciconelli RM, Morinaga LK, Breda AP, Hoette S and Souza R. Quality of life as a prognostic marker in pulmonary arterial hypertension. *Health and quality of life outcomes*. 2014;12:130.
- 120. Taichman DB, Shin J, Hud L, Archer-Chicko C, Kaplan S, Sager JS, Gallop R, Christie J, Hansen-Flaschen J and Palevsky H. Health-related quality of life in patients with pulmonary arterial hypertension. *Respiratory research*. 2005;6:92.
- 121. Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M and Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS)Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). *European heart journal*. 2015.
- 122. Ventetuolo CE, Benza RL, Peacock AJ, Zamanian RT, Badesch DB and Kawut SM. Surrogate and Combined End Points in Pulmonary Arterial Hypertension. *Proc Am Thorac Soc.* 2008;5:617-622.
- 123. ATS statement: guidelines for the six-minute walk test. *American journal of respiratory and critical care medicine*. 2002;166:111-7.
- 124. Goebelsmann U, Arce JJ, Thorneycroft IH and Mishell DR, Jr. Serum testosterone concentrations in women throughout the menstrual cycle and following HCG administration. *American journal of obstetrics and gynecology*. 1974;119:445-52.
- 125. Probst-Hensch NM, Ingles SA, Diep AT, Haile RW, Stanczyk FZ, Kolonel LN and Henderson BE. Aromatase and breast cancer susceptibility. *Endocrine-related cancer*. 1999;6:165-73.
- 126. Sodergard R, Backstrom T, Shanbhag V and Carstensen H. Calculation of free and bound fractions of testosterone and estradiol-17 beta to human plasma proteins at body temperature. *J Steroid Biochem*.

1982;16:801-10.

- 127. Vermeulen A, Verdonck L and Kaufman JM. A critical evaluation of simple methods for the estimation of free testosterone in serum. *The Journal of clinical endocrinology and metabolism*. 1999;84:3666-72.
- 128. Rinaldi S, Geay A, Dechaud H, Biessy C, Zeleniuch-Jacquotte A, Akhmedkhanov A, Shore RE, Riboli E, Toniolo P and Kaaks R. Validity of free testosterone and free estradiol determinations in serum samples from postmenopausal women by theoretical calculations. *Cancer epidemiology, biomarkers & prevention: a publication of the American Association for Cancer Research, cosponsored by the American Society of Preventive Oncology.* 2002;11:1065-71.
- 129. Rabinovitch M, Guignabert C, Humbert M and Nicolls MR. Inflammation and Immunity in the Pathogenesis of Pulmonary Arterial Hypertension. *Circulation Research*. 2014;115:165-175.
- 130. Pelletier MM, Kleinbongard P, Ringwood L, Hito R, Hunter CJ, Schechter AN, Gladwin MT and Dejam A. The measurement of blood and plasma nitrite by chemiluminescence: Pitfalls and solutions. *Free Radical Biology and Medicine*. 2006;41:541-548.
- 131. Wang X, Bryan NS, MacArthur PH, Rodriguez J, Gladwin MT and Feelisch M. Measurement of nitric oxide levels in the red cell: validation of tri-iodide-based chemiluminescence with acid-sulfanilamide pretreatment. *J Biol Chem.* 2006;281:26994-7002.
- 132. Deem S, Kim SS, Min J-H, Eveland R, Moulding J, Martyr S, Wang X, Swenson ER and Gladwin MT. Pulmonary vascular effects of red blood cells containing S-nitrosated hemoglobin. *American Journal of Physiology Heart and Circulatory Physiology*. 2004;287:H2561-H2568.
- 133. McMahon TJ, Ahearn GS, Moya MP, Gow AJ, Huang Y-CT, Luchsinger BP, Nudelman R, Yan Y, Krichman AD, Bashore TM, Califf RM, Singel DJ, Piantadosi CA, Tapson VF and Stamler JS. A nitric oxide processing defect of red blood cells created by hypoxia: Deficiency of S-nitrosohemoglobin in pulmonary hypertension. *Proceedings of the National Academy of Sciences of the United States of America*. 2005;102:14801-14806.
- 134. Skoro-Sajer N, Mittermayer F, Panzenboeck A, Bonderman D, Sadushi R, Hitsch R, Jakowitsch J, Klepetko W, Kneussl MP, Wolzt M and Lang IM. Asymmetric Dimethylarginine Is Increased in Chronic Thromboembolic Pulmonary Hypertension. *American journal of respiratory and critical care medicine*. 2007;176:1154-1160.
- 135. Kielstein JT, Bode-Böger SM, Hesse G, Martens-Lobenhoffer J, Takacs A, Fliser D and Hoeper MM. Asymmetrical Dimethylarginine in Idiopathic Pulmonary Arterial Hypertension. *Arteriosclerosis, Thrombosis, and Vascular Biology*. 2005;25:1414-1418.
- 136. Michelakis E, Tymchak W, Lien D, Webster L, Hashimoto K and Archer S. Oral Sildenafil Is an Effective and Specific Pulmonary Vasodilator in Patients With Pulmonary Arterial Hypertension: Comparison With Inhaled Nitric Oxide. *Circulation*. 2002;105:2398-2403.
- 137. Kim-Shapiro DB and Gladwin MT. Pitfalls in measuring NO bioavailability using NOx. *Nitric oxide : biology and chemistry / official journal of the Nitric Oxide Society*. 2015;44:1-2.
- 138. Rhodes P, Leone AM, Francis PL, Struthers AD, Moncada S and Rhodes PM. The L-arginine:nitric oxide pathway is the major source of plasma nitrite in fasted humans. *Biochemical and biophysical research communications*. 1995;209:590-6.
- 139. Livak KJ and Schmittgen TD. Analysis of relative gene expression data using real-time quantitative PCR and the 2(-Delta Delta C(T)) Method. *Methods (San Diego, Calif)*. 2001;25:402-8.
- 140. Gaskill C and Majka SM. A high-yield isolation and enrichment strategy for human lung microvascular endothelial cells. *Pulmonary Circulation*. 2017;7:108-116.
- 141. Bradlow WM, Hughes ML, Keenan NG, Bucciarelli-Ducci C, Assomull R, Gibbs JS and Mohiaddin RH. Measuring the heart in pulmonary arterial hypertension (PAH): implications for trial study size. *J Magn Reson Imaging*. 2010;31:117-24.
- 142. Leuchte HH, Holzapfel M, Baumgartner RA, Ding I, Neurohr C, Vogeser M, Kolbe T, Schwaiblmair M and Behr J. Clinical significance of brain natriuretic peptide in primary pulmonary hypertension. *Journal of the American College of Cardiology*. 2004;43:764-770.
- 143. Hiramoto Y, Shioyama W, Higuchi K, Arita Y, Kuroda T, Sakata Y, Nakaoka Y, Fujio Y and Yamauchi-Takihara K. Clinical significance of plasma endothelin-1 level after bosentan administration in pulmonary arterial hypertension. *Journal of Cardiology*. 53:374-380.
- 144. Lauer T, Preik M, Rassaf T, Strauer BE, Deussen A, Feelisch M and Kelm M. Plasma nitrite rather than nitrate reflects regional endothelial nitric oxide synthase activity but lacks intrinsic vasodilator action. *Proceedings of the National Academy of Sciences of the United States of America*. 2001;98:12814-9.

- 145. Kawut SM, Archer-Chicko CL, DiMichele A, Fritz JS, Klinger JR, Ky B, Palevsky HI, Palmisciano AJ, Patel M, Pinder D, Propert KJ, Smith KA, Stanczyk F, Tracy R, Vaidya A, Whittenhall ME and Ventetuolo CE. Anastrozole in Pulmonary Arterial Hypertension (AIPH): A Randomized, Double-Blind Placebo-Controlled Trial. *American journal of respiratory and critical care medicine*. 2016.
- 146. Schafer M, Kheyfets VO, Schroeder JD, Dunning J, Shandas R, Buckner JK, Browning J, Hertzberg J, Hunter KS and Fenster BE. Main pulmonary arterial wall shear stress correlates with invasive hemodynamics and stiffness in pulmonary hypertension. *Pulmonary circulation*. 2016;6:37-45.
- 147. Nilsson CG, Lahteenmaki PL, Luukkainen T, and Robertson DN. (1986). Sustained intrauterine release of levonorgestrel over five years. *Fertility and sterility*, 1986;45(6):805–807.